# A Phase III, Open-label Study of MT-6548 in Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan

## **Study Protocol**

## Study sponsor:

Mitsubishi Tanabe Pharma Corporation

Study protocol no.: MT-6548-J04

Version no.: 01.00.00000

Date: 2017/12/26

NCT number: NCT03461146

Note; This document was translated into English

from the Japanese original version.

#### CONFIDENTIALITY

This study protocol contains information which should be viewed only by those directly involved with the study. The contents of this document should only be published or disclosed to third parties with the express written consent of Mitsubishi Tanabe Pharma Corporation.

The study will be performed in compliance with the Pharmaceutical Affairs Law, Ordinance on Good Clinical Practice (GCP), related regulations, and this study protocol.

## Contents

| Protocol Summary | 1 |
|---|---|
| 1. Protocol history and background information | 15 |
| 2. Study objectives | 24 |
| 3. Subjects | 25 |
| 3.1 Subjects | 25 |
| 3.2 Inclusion criteria | 25 |
| 3.3 Exclusion criteria. | 26 |
| 3.4 Re-testing/re-screening. | 28 |
| 4. Explanations to subjects and consent | 29 |
| 4.1 Informed consent forms and written information | 29 |
| 4.2 Content of written information | 29 |
| 4.3 Method of obtaining consent | 30 |
| 4.4 Revision of informed consent forms and written information | 31 |
| 5. Study Design | 32 |
| 5.1 Study phase and type | 32 |
| 5.2 Study design | 32 |
| 5.3 Endpoints | 33 |
| 6. Target sample size and study period | 35 |
| 6.1 Target sample size | 35 |
| 6.2 Study period | 35 |
| 7. Study drug | 36 |
| 7.1 Study drug names | 36 |
| 7.2 Study drug packaging and labelling | 36 |
| 7.3 Storage method | 36 |
| 7.4 Study drug handling, storage, and management methods | 36 |
| 8. Subject-related test methods | 37 |
| 8.1 Lists of screened subjects, enrolled subjects, and identification codes | 37 |
| 8.2 Subject enrollment | 37 |
| 8.3 Dosage and administration | 38 |
| 8.4 Treatment period | 40 |
| 8.5 Concomitant medications and therapies and rescue therapy | 40 |
| 8.6 Subject oversight | 44 |
| 9. Tests and observations | 47 |
| 9.1 Test and observation schedule | 47 |
| 9.2 Test and observation timepoints | 50 |

| 10. Evaluation methods and standards | 60 |
|---|---|
| 10.1 Efficacy | 60 |
| 10.2 Safety | 62 |
| 11. Ensuring subject safety | 63 |
| 11.1 Responses to serious adverse events | 63 |
| 11.2 Significant adverse events | 63 |
| 11.3 Pregnancy reporting | 63 |
| 11.4 Contacting subjects' other doctors | 63 |
| 12. Withdrawal criteria and procedures | 65 |
| 12.1 Withdrawal criteria | 65 |
| 12.2 Procedures for withdrawal | 65 |
| 13. Statistical analysis | 67 |
| 13.1 Analysis sets | 67 |
| 13.2 Data handling | 67 |
| 13.3 Statistical analysis protocol | 68 |
| 13.4 Changes in statistical analysis protocol | 70 |
| 14. Study protocol compliance, deviation, and modification | 70 |
| 14.1 Study protocol agreement and compliance | 70 |
| 14.2 Study protocol deviations and modifications | 70 |
| 15. Revisions to the study protocol | 71 |
| 16. Termination or suspension of the entire study | 71 |
| 17. Case report forms | 72 |
| 17.1 Case report form (CRF) format | 72 |
| 17.2 Direct recording of information in the CRF and CRF as source documents | 72 |
| 17.3 Notes on making CRF entries | 73 |
| 17.4 CRF submission timepoints | 73 |
| 18. Direct access to source documents | 74 |
| 19. Study quality control and quality assurance | 74 |
| 20. Ethics | 74 |
| 20.1 Ethical conduct of the study | 74 |
| 20.2 Institutional Review Board. | 74 |
| 20.3 Subject confidentiality | 75 |
| 21. Record storage | 75 |
| 22. Monetary compensation | 75 |
| 23. Compensation for health damage and insurance | 76 |
| 23.1 Compensation for health damage | 76 |
| 23.2 Insurance | 76 |

| 24. Publication policy | ) |
|-------------------------------------------------------------|----------|
| 25. Genetic analysis study | ŗ |
| 25.1 Purpose of the study | ! |
| 25.2 Eligible subjects | , |
| 25.3 Obtaining consent | , |
| 25.4 Sample handling77 | , |
| 25.5 Performing genetic analysis | í |
| 25.6 Publication of results and disclosure to sample donors | <b>;</b> |
| 26. Administrative structure | , |
| <b>26.1</b> Study sponsor: | ÷ |
| 26.2 Study centers and investigators | , |
| 27. References 81 | |
| Accompanying documents | |
| Attachment 1 Pregnancy Reports | |
| Appendices | |
| Appendix 1 Administrative structure | |
| Appendix 2 List of Study centers and investigators | |
| Appendix 3 Study protocol agreement | |
| Appendix 4 EQ-5D-5L questionnaires | |
| Appendix 5 KDQOL questionnaires | |

#### List of abbreviations

| Abbreviation | |
|---|---|
| AUC | Area under the plasma concentration-time curve |
| BCRP | Breast cancer resistance protein |
| CKD | Chronic kidney disease |
| | Maximum plasma concentration |
| C <sub>max</sub><br>CYP | Cytochrome P450 |
| DNA | Deoxyribonucleic acid |
| DIVA | Electronic data capture: Systems for using electronic devices and software to collect |
| EDC | data on clinical study subjects from study centers or contract testing laboratories |
| EPO | Erythropoietin |
| ESA | Erythropoiesis stimulating agent |
| FAS | Full analysis set |
| GFR | Glomerular filtration rate |
| GCP | Good clinical practice |
| HD-CKD | Hemodialysis dependent chronic kidney disease |
| HIF-PH | Hypoxia inducible factor prolyl hydroxylase |
| IC <sub>50</sub> | Median inhibitory concentration |
| JSDT | The Japanese society for dialysis therapy |
| LOCF | Last observation carried forward |
| MMRM | Mixed model repeated measures |
| MRP | Multidrug resistance-associated protein |
| NDD-CKD | Nondialysis dependent chronic kidney disease |
| OATP | Organic anion transporting polypeptide |
| OAT | Organic anion transporter |
| PD | Pharmacodynamics |
| P-gp | P-glycoprotein |
| PK | Pharmacokinetics |
| PT | Preferred term |
| QOL | Quality of life |
| SOC | System organ class |
| t <sub>1/2</sub> | Terminal elimination half-life |
| $T_{\text{max}}$ | Time to reach maximum plasma concentration |
| TIBC | Total iron binding capacity |
| TSAT | Transferrin saturation |

### Definitions of Terms

| Term | Definitions |
|---|---|
| Study period | From the day of informed consent to the final day of |
| | follow-up observation period |
| Treatment period | From the first day of the treatment period to the final day of |
| | the treatment period |
| Day of completion of treatment period | Week 24 of treatment period or day of discontinuation of |
| | treatment |
| X weeks prior to the first day of the | Same day of week from X weeks prior to the first day of the |
| screening period. | screening period |
| MT-6548 Tablet | Each film-coated tablet contains 150 mg vadadustat. |

#### **Protocol Summary**

#### 1. Study title

A phase III, open-label study of MT-6548 in hemodialysis subjects with anemia associated with chronic kidney disease in Japan

#### 2. Purpose of the study

The study will evaluate the effects of MT-6548 on improvement and maintence in hemoblobin (Hb) levels and safety in patients with anemia associated with hemodialysis-dependent chronic kidney disease (HD-CKD) who are not corrently treated with any erythropoiesis-stimulating agent (ESA).

#### 3. Subjects

#### 3.1 Subjects

Patients with anemia associated with HD-CKD

#### 3.2 Inclusion criteria

Subjects must meet all inclusion criteria below and have capacity to grant informed consent. Laboratory tests related to the inclusion criteria will be assessed based on central laboratory measurements. If a given laboratory test is performed multiple times during the screening period, the most recent test will be used for assessment. If blood is drawn on the day of dialysis, data obtained before dialysis will be used for assessment. In addition, Hb values in blood collected in the supine position will be used for assessment.

- (1) Patients at least 20 years of age as of the day of consent (either sex)
- (2) Patients with CKD diagnosed according to the Japanese Society of Nephrology's "Clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012" as of the day of consent
- (3) Patients who have received either hemodialysis or hemodiafiltration three times a week however, patients on home dialysis and those receiving a combined therapy of home hemodialysis and peritoneal dialysis are excluded
- (4) Patients who have not received any ESA formulation for at least the following period prior to the first day of the screening period; however, patients who have received ESA formulations should discontinue administration after giving informed consent and undergo a washout of at least the following period prior to the first day of the screening period.
  - ✓ Epoetin alpha (recombinant), epoetin beta (recombinant), and epoetin kappa (recombinant): 1 week
  - ✓ Darbepoetin alfa (recombinant): 2 weeks
  - ✓ Epoetin beta pegol (recombinant): 4 weeks

- (5) Patients with a mean Hb value (mean of the latest two measurements) of ≥8.0 g/dL and <10.0 g/dL during the screening period
- (6) Patients with an Hb difference of <1.5 g/dL between the latest two measurements during the screening period
- (7) Patients with a serum ferritin value of ≥100 ng/mL or a transferrin saturation (TSAT) of ≥20% during the screening period
- (8) Patients with folic acid and vitamin B<sub>12</sub> values above the lower limit of normal values during the screening period

#### 3.3 Exclusion criteria

Patients who meet any of the following exclusion criteria will be excluded. Laboratory tests related to the exclusion criteria will be assessed based on central laboratory measurements. If a given laboratory test is performed multiple times during the screening period, the most recent test will be used for assessment. If blood is drawn on the day of dialysis, data before dialysis will be used for assessment.

- (1) Patients who have anemia primarily due to diseases other than CKD (including sickle cell disease, myelodysplastic syndrome, myelofibrosis, hematopoietic malignancy, myeloma, hemolytic anemia, thalassemia, and pure red cell aplasia) after the day of informed consent
- (2) Patients with active haemorrhaging or exsanguination within 8 weeks prior to the first day of the screening period
- (3) Patients who have received RBC transfusion within 8 weeks prior to the first day of the screening period
- (4) Patients who have received testosterone enanthate or mepitiostane within 8 weeks prior to the first day of the screening period
- (5) Patients determined by investigators/subinvestigators to likely require immediate rescue therapy or drug holiday of the study drug after initiation of treatment period
- (6) Patients who are expected to no longer require hemodialysis or hemodiafiltration due to recovery of renal function
- (7) Patients with AST, ALT, or total bilirubin values of 2.5 times or greater the upper limit of standard during the screening period. This does not apply to patients with Gilbert's syndrome.
- (8) Patients with poorly controlled hypertension (defined as a systolic blood pressure (BP) of >180 mmHg or diastolic BP of >110 mmHg) on the first day of the screening period and on the first day of the treatment period
- (9) Patients for whom any of the following apply upon fundoscopy during the screening period:
  - ✓ No ocular fundus findings are possible.
  - ✓ Active ocular fundus disease

- (10) Patients with severe cardiac failure from the day of consent (Class IV according according to severity classification of the New York Heart Association [NYHA])
- (11) Patients with cerebrovascular disorders or acute coronary syndromes (hospitalization for unstable angina or myocardial infarction, etc.) within 12 weeks prior to the first day of the screening period. Patients who have been hospitalized due to acute coronary angioplasty or cardiac failure.
- (12) Patients with malignant tumors or a history of such. However, this does not apply to patients with no relapse for 5 or more years (5 or more years with no relapse from last administration of chemotherapy if chemotherapy was used).
- (13) Patients with incidence or relapse of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the first day of the screening period
- (14) Patients with current or previous haemosiderosis or hemochromatosis
- (15) Patients with a history of or plans for organ transplant (not including being on a waiting list for renal transplant), haematopoietic stem cell transplant, or bone marrow transplant
- (16) Patients with an allergy to the study drugs
- (17) Patients who have participated in another clinical study and received study drugs within 12 weeks prior to informed consent, or within 5 times the half-life of the study drug (whichever is longer)
- (18) Patients who have previously used MT-6548
- (19) Patients who are known not to be tolerant to hypoxia-inducible factor prolyl hydroxylase enzyme inhibitors
- (20) Patients who are unwilling to consent to use contraception from the beginning of the study period to 30 days following the final dose of the study drug for women who may become pregnant, or from the beginning of the study period to 90 days following the final dose of the study drug for men
- (21) Female patients who are or may be pregnant, or women who are nursing
- (22) Other patients judged by investigators/subinvestigators to be inappropriate as a subject in this study

#### 3.4 Re-testing/re-screening

#### (1) Re-testing

Re-testing may be performed during the screening period at the discretion of the investigator/subinvestigator for any subject whose laboratory values (Hb, serum ferritin, TSAT, folic acid, vitamin B<sub>12</sub>, AST, ALT, and total bilirubin) or BP do not meet the inclusion criteria or meet the exclusion criteria during the screening period.

Subjects with blood pressure measurements on the first day of the treatment period which meet exclusion criteria may be re-tested at the discretion of investigators/subinvestigators, and processed for treatment period initiation if they no longer meet exclusion criteria.

However, the maximum time from the first day of the screening period to the first day of the treatment period is 6 weeks.

#### (2) Re-screening

For any subject whose laboratory values (Hb, serum ferritin, TSAT, folic acid, vitamin B<sub>12</sub>, AST, ALT, and total bilirubin), BP, or BP measurements on the first day of the treatment period do not meet the inclusion criteria or meet the exclusion criteria during the screening period, re-screening may be performed if the investigator/subinvestigator considers that the subject may become eligible for the study due to natural course or with drug therapy.

However, re-screening may only be performed once for any given subject.

#### 4. Study design

This is a multicenter, uncontrolled, open-label study.



#### (1) Screening period

The screening period begins on the first day of the screening period, and ends upon completion of tests required on the first day of the treatment period. Maximum screening period time is 6 weeks. Two visits will be made during the screening period; the first (SV1) is the first day of the screening period. The second screening period visit (SV2) occurs after results from laboratory tests performed on the first day of the screening period have been obtained. Testing may be repeated as necessary.

#### (2) Treatment period

The treatment period will last from completion of scheduled tests on the first day of the treatment period to completion of blood sampling for haematology tests on the final day of the treatment period (Week 24 of the treatment period or discontinuation of treatment).

During the treatment period, subjects are to visit the study site on the day of dialysis after a 2-day interdialytic interval; however, if this is difficult, subjects are to visit the study site on the day of dialysis after a 1-day interdialytic interval. After the first day of the treatment period, subjects are to visit the study site every 2 weeks until Week 12 and every 4 weeks after Week 12 to undergo the scheduled test. However, subjects are to visit the study site at shorter intervals as necessary, if excessive increases or decreases in Hb are of concern based on the time course of Hb levels or for hemodialysis.

#### (3) Follow-up observation period

The follow-up observation period consists of 2 weeks from completion of blood sampling for haematology tests on the final day of the treatment period. The final day of the follow-up observation period is 2 weeks from the completion of blood sampling for haematology tests on the final day of the treatment period, regardless of whether a study visit is made on that day.

Subjects should make study visits as close to the same time as possible during the study period for scheduled tests.

5. Study drug, dosage, and administration

5.1 Study drug name

Name: MT-6548 Tablet 150 mg Nonproprietary name: vadadustat

Dosage form and content: Each film-coated tablet contains 150 mg vadadustat.

5.2 Dosage and administration

5.2.1 Initial dose

Single daily dose of 300 mg (2 tablets)

5.2.2 Maintenance dosage and dosage adjustments

Maintenance dosage is 150-600 mg once daily and adjusted according to the dosage adjustment guideline below.

[MT-6548 Tablet dosage adjustment guidelines]

Investigators/subinvestigators will monitor Hb levels throughout the treatment period, and determine whether to adjust study drug dosage or discontinue administration as required. In principle, dosage adjustments should be performed at scheduled visits; however, an unscheduled visit may be provided for dosage adjustment, if considered necessary, in cases where excessive increases or decreases in Hb levels are of concern based on the Hb time course.

Hb levels will be measured in samples collected in the supine position using a HemoCue<sup>®</sup> Hb201 DM analyzer; and in principle, these measurements will be used to determine dosage adjustments. Hb levels on the day of dialysis will be measured in samples collected before dialysis. Hb measurements used for dosage adjustment determinations will be recorded in the subject's CRF. Measurement results from the HemoCue<sup>®</sup> Hb201 DM will be used solely for determination of study drug dosage adjustments, and will not be used for efficacy or safety analysis.

The dosage adjustment algorithm below will be followed in order to improve and maintain Hb levels of 10.0–12.0 g/dL during the study. Dosage steps are defined in the dosage adjustment table below.

6

MT-6548 Tablet dosage adjustment table

| Step | No. of tablets | Dosage |
|------|----------------|--------|
| 1 | 1 | 150 mg |
| 2 | 2 | 300 mg |
| 3 | 3 | 450 mg |
| 4 | 4 | 600 mg |

\*It is permitted for dosage adjustments not to comply with the dosage adjustment algorithm for safety reasons depending on factors such as clinical status (e.g., AEs, volume depletion, or volume overload), Hb elevation rate, decrease rate, or fluctuations. In such cases, clinical status will be recorded in CRFs. All dosage increases of MT-6548 will be in increments of 1 tablet at a time.

If a dosage increase or reduction according to the dosage adjustment algorithm is impossible because the maximum or minimum dosage on the dosage adjustment table is already being administered, it is permitted to not alter the dosage at that point. However, in this case it will be confirmed whether withdrawal criteria are met, and treatment discontinued if so.

#### MT-6548 Tablet dosage adjustment algorithm

- ✓ Dosage increases should be performed at intervals of at least 4 weeks in principle, and dosage decreases at intervals of at least 2 weeks.
- ✓ If Hb levels suddenly increase (>2.0 g/dL change in the past 4 weeks\*), decrease MT-6548 dosage by 1 tablet.
- ✓ Increase MT-6548 dosage by 1 tablet if Hb levels are <10.0 g/dL. However, decrease by 1 tablet instead of increasing in cases of sudden increase in Hb (more than 2.0 g/dL change in past 4 weeks\*).
- ✓ Decrease MT-6548 dosage by 1 tablet if Hb levels are >11.5 g/dL.
- ✓ If Hb levels are >12.0 g/dL and ≤13.0 g/dL with a rapid increase in Hb levels (>2.0 g/dL change in the past 4 weeks\*), MT-6548 tablet administration should be discontinued, and the dose should be decreased by 1 tablet and MT-6548 tablet administration resumed after Hb levels decrease to ≤12.0 g/dL.
- ✓ If Hb levels are >13.0 g/dL, MT-6548 tablet administration should be discontinued, and the dose should be decreased by 1 tablet and MT-6548 tablet administration resumed after Hb levels decrease to ≤12.0 g/dL.

\*The rate of increase in Hb levels will be calculated using the Hb levels at the time points closest to 4 weeks among those measured 3–5 weeks prior to the day of dosage adjustment. A rate of change greater than 0.5 g/dL/week will be regarded as a rapid increase in Hb

levels. If no Hb levels were measured 3–5 weeks prior to the day of dosage adjustment, the Hb levels measured at most recent time points prior to 5 weeks before the day of dosage adjustment will be used to calculate the rate of increase in Hb levels.

#### 5.2.3 Administration method

The study drug is taken once-daily orally. The drug does not need to be taken with meals, but timing should be as consistent as possible throughout the treatment period, both in relation to meals and time of day. (The first dose will be taken after required tests are finished on the first day of the treatment period.)

#### 5.3 Duration of treatment

From the first day of the treatment period to the day before Week 24 of the treatment period

#### 6. Concomitant medications/therapies and rescue therapy

#### 6.1 Prohibited concomitant medications and therapies

#### (1) ESA formulations

Concomitant use of ESA formulations is prohibited during the following period. These restrictions do not apply to rescue therapy.

- 1) Epoetin alpha (recombinant), epoetin beta (recombinant), and epoetin kappa (recombinant): from 1 week prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.
- 2) Darbepoetin alfa (recombinant): from 2 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.
- 3) Epoetin beta pegol (recombinant): from 4 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.

#### (2) Testosterone enanthate and mepitiostane

Concomitant use is prohibited from 8 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.

#### (3) Blood transfusion

Prohibited from 8 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. These restrictions do not apply to rescue therapy.

#### 6.2 Restricted concomitant medications and therapies

#### (1) Iron supplements

From the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period, administer iron supplements to maintain serum ferritin values of  $\geq 100$  ng/mL or TSAT of  $\geq 20\%$ . Iron supplements may be omitted for subjects who respond poorly to them, such as those with an allergy or those with adverse drug reaction (ADRs) to iron (vomiting, etc.).

Investigators/subinvestigators will determine iron supplement dosage and administration route.

Important: Oral iron supplements may impair MT-6548 bioavailability, so oral iron supplements must not be taken at the same time as MT-6548 Tablet. Subjects taking oral iron supplements will be instructed not to take any within 2 hours before or after taking MT-6548 Tablet.

#### (2) Iron-containing phosphate binders (ferric citrate hydrate, sucroferric oxyhydroxide)

New use of iron-containing phosphate binders is fundamentally prohibited from the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. If iron-containing phosphate binders are used by a subject on the first day of the screening period, then the same dosage of the same type should fundamentally be continued from the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. If investigators/subinvestigators determine that a dosage increase is required for iron-containing phosphate binders, then additional treatment will be performed with hyperphosphatemia drugs containing no iron, or treatment switched to hyperphosphatemia drugs containing no iron. Dosage of iron-containing phosphate binders may also be reduced if determined necessary according to the subject's condition. Switching to another hyperphosphatemia drug containing no iron will not be permitted during the period from the first day of the screening period to completion of designated tests for treatment period Week 4.

Important: As with oral iron supplements, iron-containing phosphate binders may impair MT-6548 bioavailability, so iron-containing phosphate binders must not be taken at the same time as MT-6548 Tablet. Subjects taking iron-containing phosphate binders will be instructed not to take any within 2 hours before or after taking MT-6548 Tablet.

#### (3) Hemodialysis

The type of hemodialysis is either hemodialysis or hemodiafiltration with a frequency of

three times a week. In principle, a change in the type and frequency of hemodialysis is prohibited from the first day of the screening period to the completion of blood sampling for hematology tests on the final day of the treatment period; however, the type (hemodialysis and hemodiafiltration) and frequency may be changed if the investigator/subinvestigator considers it clinically necessary.

#### 6.3 Rescue therapy

The following rescue therapy options will be provided as needed for subject safety. Even if rescue therapies are performed, the subject can continue in the study unless investigators/subinvestigators determine study withdrawal is appropriate. Details of any rescue therapy implemented will be recorded in the subject's CRF.

#### (1) ESA formulations

If a subject has received maximum dosages of MT-6548 Tablets for ≥2 weeks and meets all criteria below, the investigator/subinvestigator may administer an ESA as a rescue therapy to improve Hb levels if necessary in order to secure subject safety. An ESA-based rescue therapy may also be provided without meeting the criteria below if the investigator/subinvestigator considers it necessary to secure subject safety, such as in cases of acute decreases in Hb levels. MT-6548 Tablets administration will be discontinued when an ESA-based rescue therapy is provided. MT-6548 Tablets administration may be resumed after an improvement in Hb levels and should not be coadministered with a rescue therapy with an ESA. Subjects who are not expected to resume MT-6548 Tablets administration will be withdrawn from the study.

- ✓ Anaemia or anaemia symptoms (e.g., fatigue, weakness, shortness of breath, chest pain, confusion, dizziness) become aggravated compared to the first day of the treatment period to the point they are clinically problematic.
- ✓ Hb levels drop to <8.0 g/dL.

#### (2) RBC transfusion

Usually, RBC transfusions are performed when clinically necessary in instances of acute or major bleeding. For less sever anemia, which may be exacerbated, or moderate to severe anemia symptoms, RBC transfusions may be performed as needed clinically at the discretion of the investigator/subinvestigator.

#### (3) Phlebotomy

Phlebotomy may be performed at investigator/subinvestigator discretion in cases of hyperviscosity syndrome, if the rate of Hb increase is concerning to

investigators/subinvestigators, or if Hb levels are high enough to warrant concern to investigators/subinvestigators.

#### 7. Endpoints

#### 7.1 Efficacy endpoints

- (1) Primary endpoint
  - 1) Mean Hb at treatment period Weeks 20 and 24
  - 2) Hb at each treatment period timepoint
  - 3) Proportion of subjects with mean Hb levels within the target range (10.0–12.0 g/dL), <10.0 g/dL, and  $\ge$ 12.0 g/dL at each timepoint in the treatment period
  - 4) Number of days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL)
  - 5) Rate of increase in Hb levels

#### (2) Other endpoints

- 1) Change in mean Hb at treatment period Weeks 20 and 24
- 2) Proportion of subjects with a ≥1.0 g/dL increase from baseline in mean Hb levels at Weeks 20 and 24 of the treatment period
- 3) Ratio of subjects who received ESA rescue therapy
- 4) Ratio of subjects who received red blood cell (RBC) transfusion rescue therapy.
- 5) Study drug dosage
- 6) Total number of study drug dosage adjustments
- 7) Quantity of iron administered
- 8) Ratio of subjects with serum ferritin of  $\geq$ 100 ng/mL or TSAT  $\geq$ 20%.
- 9) Change from baseline of iron-related measures (serum iron, total iron binding capacity (TIBC), TSAT, and serum ferritin) and hepcidin.
- 10) Changes from baseline in haematocrit, RBC count, reticulocytes (count and fraction), and erythropoietin (EPO)
- 11) QOL measures (EQ-5D-5L, KDQOL)

#### 7.2 Safety endpoints

- (1) Adverse events and adverse drug reactions
- (2) Laboratory test values
- (3) Resting standard 12-lead ECG
- (4) Dry weight
- (5) Body weight
- (6) Vital signs
- (7) Fundoscopy

- (8) Chest X-ray
- (9) Proportion of subjects with documented Hb levels of ≥12.0 or ≥13.0 g/dL
- (10) Ratio of subjects with Hb increase rates exceeding 0.5 g/dL/week.

#### 8. Withdrawal criteria

Subjects will be withdrawn from the study if the following criteria are met:

- (1) If the subject expresses a desire to withdraw from the study.
- (2) If it is discovered that the subject is clearly ineligible for study participation.
- (3) If investigators/subinvestigators determine that AEs make continued participation in the study difficult.
- (4) If investigators/subinvestigators determine that continuation of the study is inappropriate for a subject, such as if hyperviscosity syndrome occurs or if control of Hb within the target range is impossible.
- (5) If the subject no longer requires hemodialysis or hemodiafiltration.
- (6) If the subject has undergone renal transplantation.
- (7) If pregnancy of the subject is discovered.
- (8) If the investigator/subinvestigator determines a subject should withdraw from the study for any other reason.

#### 9. Target sample size

The number of subjects registered in the treatment period will be 20.

#### 9.1 Rationale for target sample size

The proportion of patients who are not treated with any ESA formulation is as small as approximately 10% of all hemodialysis-dependent patients in Japan. Patients receiving any ESA formulation are allowed to register after undergoing a washout; however, the number of eligible patients was thought to be very limited when considering the selection/exclution criteria. Therefore, the target sample size was set to 20 after consideration of feasibility.

#### 10. Study period

11. Test and observation schedule

| | | | | | | | | | - | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| / | | Screening period [a] | period [a] | | | | | Ĭ | I reatment period [b] | riod [b] | | | | | Final day of |
| Visit | Informed | First day | Visit 2 | First day<br>[b] | W2 | W4 | W6 | W8 | W10 | W12 | W16 | W20 | W24 | Day of discontinuation | the follow-up<br>observation [c] |
| Visit number | ıc | IAS | ZAS | IVI | TVZ | TV3 | TV4 | TV5 | TV6 | TV7 | TV8 | TV9 | TV10 | TV11 | FU |
| Permitted range (days) | - | - | , | - | #3 | #3 | #3 | ∓3 | ∓3 | ∓3 | <b>L</b> ∓ | <b>L</b> ∓ | +7 | +7 or +14 [e] | +7 |
| Procedure/evaluation | | | | | | | | | | | | | | | |
| Informed consent | x | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | × | х | х | х | | | | | | | | | | | |
| Patient backgroud and history | × | | | х | | | | | | | | | | | |
| Height | | | | х | | | | | | | | | | | |
| Dry weight, body weight [f] | | | | х | | | | | | × | | | × | Х | |
| Folic acid and vitamin $B_{12}$ [g] | | X | | | | | | | | | | | | | |
| Pregnancy tests [i] | | Х | | | | | | | | | | | × | Х | |
| Hematology tests [g], [h], [j] | | × | X [k] | х | х | х | х | х | x | х | х | x | × | Х | |
| Blood biochemistry tests [g], [h], [l] | | Х | | Х | х | x | x | × | x | × | × | x | × | X | |
| C-reactive protein [g], [h] | | х | | × | | | | | | | | | × | × | |
| Ion-related measures [g], [h] | | × | | × | × | × | × | × | × | × | × | × | × | × | |
| Hepcidin [h] | | | | × | × | × | × | | | × | | | × | X | |
| EPO [h] | | | | × | × | × | × | | | × | | | × | × | |
| VEC#[h] | | | | × | | | | | | × | | | × | Х | |
| Vital signs [g], [h], [m] | | х | | Х | х | x | х | × | x | x | х | x | × | × | |
| Resting standard 12-lead ECG [h], [n] | | | | x | | | | | | | | | × | Х | |
| Fundoscopy [e] | | ζ. | x | | | | | | | | | × | Ĵ | X | |
| Chest X-ray [e] | | ۲ | x | | | | | | | | | × | Ţ | × | |
| Duration of hemodialysis | | | | × | | | | | | | | | × | × | |
| QOL measures (EQ-5D-5L, KDQOL) | | | | × | | | | | | X. | | | × | × | |
| AE investigation | | | | × | × | × | × | × | × | × | × | × | x | X | × |
| Blood sampling for genetic analysis [o] | | | | | Blood | Blood sampling for genetic analysis performed once as early as possible after Week 2 of treatment period | or genetic s | analysis per | formed onc | e as early a | s possible a | fter Week | 2 of treatm | ent period | |
| Product evaluation/procedure | | | | | | | | | | | | | | | |
| Investigation of concomitant medications/therapies | | | | × | х | × | х | х | x | × | × | × | х | × | × |
| MT-6548 tablets [p], [q] | | | | | | | Administer | Administered according to the dosage adjustment guidelines | ig to the do | sage adjustr | nent guidel | ines | | | |
| Iron supplements | | | | Iron sup | plements a | Iron supplements administered to maintain serum ferritin values of ≥100 ng/mL or TSAT of ≥20% | to maintai | n serum fer | ritin values | of≥100 ng | /mL or TS | AT of ≥20% | % | | |

- [a] Maximum screening period length is 6 weeks. Test results will be reviewed prior to transitioning from the first day of the screening period to screening period Visit 2, and from screening period Visit 2 to the first day of the treatment period. Re-testing will be performed as necessary.
- [b] During the treatment period, subjects are to visit the study site on the day of dialysis after a 2-day interdialytic interval; however, if this is difficult, subjects are to visit the study site on the day of dialysis after a 1-day interdialytic interval.
- [c] Not required if withdrawn prior to the treatment period.
- [d] To be performed prior to the study drug treatment (AE investigation begins after study drug administration)
- [e] Fundoscopy and chest X-ray performed once during screening period, once during Weeks 20–24 of treatment period. In the case of discontinuation of the treatment period, fundoscopy and chest X-ray should be performed within 14 days after discontinuation whenever possible.
- [f] Body weights should be measured before and after dialysis.
- [g] To be measured before dialysis on the day of dialysis during the screening period.
- [h] Tests during the treatment period should be performed before dialysis on the day of dialysis.
- [i] To be performed only in female subjects of childbearing potential.
- [j] Hb levels should be measured in blood collected in the supine position.
- [k] Only Hb levels should be measured.
- [1] Only urea nitrogen levels should be measured before and after dialysis on the first day, Week 24 of the treatment period, and on the day of treatment discontinuation.
- [m] To be measured in the sitting position after a 5-minute rest before blood sampling whenever possible.
- [n] To be measured in the supine position after a 5-minute rest before blood sampling whenever possible.
- [o] For subjects giving consent to blood sampling for genetic analysis, blood will be collected once as early as possible after Week 2 of the treatment period.
- [p] MT-6548 Tablets should be prescribed depending on the number of unused tablets by the subject. Subjects should be instructed to open a new bottle after using up the tablets in one bottle.
- [q] In principle, dosage adjustments should be performed at scheduled visits; however, an unscheduled visit may be provided for dosage adjustment, if considered necessary, in cases where excessive increases or decreases in Hb levels are of concern based on the Hb time course.

#### 1. Protocol history and background information

#### (1) Target disease and treatment methods

Chronic kidney disease (CKD) is defined in Japanese Society of Nephrology's "Clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012" as renal disorders (e.g., proteinuria) or renal impairment with glomerular filtration rate (GFR) of <60 mL/min/1.73m<sup>2</sup> for 3 or more months.

CKD is a significant public health problem throughout the world, and in Japan alone 20% of adults are estimated2) to have GFR of <60 mL/min/1.73m<sup>2</sup>. In Japan there are more than 300,000 CKD patients requiring dialysis, a number which has increased in the past 30 years<sup>3)</sup>.

Anaemia is a well-known complication of renal disease, and occurs early after onset of CKD<sup>4)</sup>. Prevalence of anaemia increases as CKD progresses, with 53% to 89% of dialysis patients affected by the disease<sup>5, 6)</sup>. Causes of anaemia in CKD patients include exsanguination, reduced RBC (red blood cell) lifespan, iron deficiency, erythropoietin (EPO) deficiency, The primary cause of nephrogenic anaemia is EPO deficiency, which results from hypoxic disorders or cells surrounding renal tubules or cell decrease in cells surrounding renal tubules<sup>4, 7)</sup>.

Further, iron loss due to dialysis is an extremely important cause of anaemia in CKD and requires iron supplementation<sup>7)</sup>. Anaemia significantly affects organ function by decreasing oxygen transport to tissue, resulting in various symptoms such as fatigue, shortness of breath, and exercise intolerance<sup>6)</sup>. Compensatory changes occur in the structure and function of the heart in these anaemia patients, including increased cardiac output and left ventricular hypertrophy, which can ultimately result in cardiac failure<sup>8)</sup>. Other anaemia-related disorders observed in CKD patients include cognitive function disorders, sleep disorders, and impaired immune function, sometimes resulting in reduced quality of life (QOL)<sup>4,9)</sup>. Anaemia is also a factor related to poor prognosis in CKD patients<sup>4,7)</sup>. Improving anaemia results particularly in markedly improved QOL in terms of energy, fatigue, and physical function<sup>4,7,10)</sup>.

Dialysis is the most popular treatment for end-stage renal disease in Japan, and hemodialysis and hemodiafiltration are particularly common modalities. A survey by the Japanese Society for Dialysis Therapy (JSDT) ("An overview of regular dialysis treatment in Japan as of December 31, 2015") showed that 79.5% of all patients on dialysis at the end of 2015 were on hemodialysis, and 17.0% were on hemodiafiltration.

Erythropoiesis-stimulating agents (ESAs), which include epoetin alfa (recombinant), epoetin beta (recombinant), epoetin kappa (recombinant), darbepoetin alfa (recombinant), and epoetin beta pegol (recombinant), are the standard therapy for anemia in patients with hemodialysis-dependent chronic kidney disease (HD-CKD).

#### (2) Study drug names and explanations

MT-6548 is a hypoxia-inducible factor prolyl hydroxylase enzyme (HIF-PH) inhibitor currently under development for treatment of anaemia in CKD patients either using or not using dialysis. It is a novel small-molecule compound which can be taken orally.

HIF-PH causes hydroxylation of HIF- $\alpha$  in normoxic conditions, reducing HIF- $\alpha$  levels with von Hippel-Lindau (VHL)-dependent breakdown of HIF- $\alpha$ . However, in hypoxic conditions HIF-PH activity is reduced, causing stabilized HIF- $\alpha$  to be transported to the cellular nucleus, where it forms a dimer with HIF- $\beta$  and binds with hypoxia response elements (HRE) to control various target genes, such as activation of EPO genes which increase EPO protein production. By inhibiting HIF-PH activity, MT-6548 creates a physiological response similar to that of hypoxic conditions, thereby increasing EPO protein production are resulting in increased Hb and RBC production<sup>11)</sup>.

(3) Nonclinical and clinical study results

Refer to the latest MT-6548 investigator's brochure for details.















#### (4) Investigational plan

The current study will evaluate efficacy and safety of MT-6548 in patients with HD-CKD-related anaemia who are not receiving ESA treatment.

Based on results of clinical studies to date, the treatment period is set at 24 weeks an appropriate period to enable evaluation of MT-6548 efficacy in terms of Hb improvement and maintenance.

MT-6548 dosage is set based on results to date at an initial dosage of 300 mg, with

maintenance dosages of 150-600 mg.

## 2. Study objectives

The study will evaluate the effects of MT-6548 on improvement and maintence in hemoblobin (Hb) levels and safety in patients with anemia associated with hemodialysis-dependent chronic kidney disease (HD-CKD) who are not corrently treated with any erythropoiesis-stimulating agent (ESA).

#### 3. Subjects

#### 3.1 Subjects

Patients with anemia associated with HD-CKD

#### 3.2 Inclusion criteria

Subjects must meet all inclusion criteria below and have capacity to grant informed consent. Laboratory tests related to the inclusion criteria will be assessed based on central laboratory measurements. If a given laboratory test is performed multiple times during the screening period, the most recent test will be used for assessment. If blood is drawn on the day of dialysis, data obtained before dialysis will be used for assessment. In addition, Hb values in blood collected in the supine position will be used for assessment.

- (1) Patients at least 20 years of age as of the day of consent (either sex)
- (2) Patients with CKD diagnosed according to the Japanese Society of Nephrology's "Clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012" as of the day of consent
- (3) Patients who have received either hemodialysis or hemodiafiltration three times a week however, patients on home dialysis and those receiving a combined therapy of home hemodialysis and peritoneal dialysis are excluded
- (4) Patients who have not received any ESA formulation for at least the following period prior to the first day of the screening period; however, patients who have received ESA formulations should discontinue administration after giving informed consent and undergo a washout of at least the following period prior to the first day of the screening period.
  - ✓ Epoetin alpha (recombinant), epoetin beta (recombinant), and epoetin kappa (recombinant): 1 week
  - ✓ Darbepoetin alfa (recombinant): 2 weeks
  - ✓ Epoetin beta pegol (recombinant): 4 weeks
- (5) Patients with a mean Hb value (mean of the latest two measurements) of ≥8.0 g/dL and <10.0 g/dL during the screening period
- (6) Patients with an Hb difference of <1.5 g/dL between the latest two measurements during the screening period
- (7) Patients with a serum ferritin value of ≥100 ng/mL or a transferrin saturation (TSAT) of ≥20% during the screening period
- (8) Patients with folic acid and vitamin B<sub>12</sub> values above the lower limit of normal values during the screening period

#### Rationale

- (1) Individuals are legally capable of granting consent as of 20 years of age. There is no particular basis for limiting participation to either sex.
- (2) To ensure that subjects have the target disease of CKD.
- (3) Set to ensure patients on hemodialysis or hemodiafiltration.
- (4) Set to ensure HD-CKD patients not being treated with an ESA formulation. Washout period set with consideration to patient safety.
- (5) Criteria set with reference to target Hb values in nephrogenic anaemia therapy according to JSDT's "Guideline for Renal Anemia in Chronic Kidney Disease 2015."
- (6) Set to ensure appropriate efficacy evaluation by targeting patients without significant fluctuations in Hb levels.
- (7) Set to ensure patients without iron insufficiency, using as reference criteria for initiating iron supplementation therapy according to the JSDT's "Guideline for Renal Anemia in Chronic Kidney Disease 2015."
- (8) Set to ensure appropriate efficacy evaluation by targeting patients without insufficiencies in folic acid or vitamin B<sub>12</sub>, required for hematopoiesis.

#### 3.3 Exclusion criteria

Patients who meet any of the following exclusion criteria will be excluded. Laboratory tests related to the exclusion criteria will be assessed based on central laboratory measurements. If a given laboratory test is performed multiple times during the screening period, the most recent test will be used for assessment. If blood is drawn on the day of dialysis, data before dialysis will be used for assessment.

- (1) Patients with anaemia resulting primarily from a disease other than CKD after date of consent (e.g., sickle-cell syndrome, myelodysplastic syndrome, myelofibrosis, haematopoietic malignancy, myeloma, haemolytic anaemia, thalassemia, or aplasia pure red cell)
- (2) Patients with active haemorrhaging or exsanguination within 8 weeks prior to the first day of the screening period
- (3) Patients who have received RBC transfusion within 8 weeks prior to the first day of the screening period
- (4) Patients who have received testosterone enanthate or mepitiostane within 8 weeks prior to the first day of the screening period
- (5) Patients determined by investigators/subinvestigators to likely require immediate rescue therapy or drug holiday of the study drug after initiation of treatment period

- (6) Patients who are expected to no longer require hemodialysis or hemodiafiltration due to recovery of renal function
- (7) Patients with AST, ALT, or total bilirubin values of 2.5 times or greater the upper limit of standard during the screening period. This does not apply to patients with Gilbert's syndrome.
- (8) Patients with poorly controlled hypertension (defined as a systolic blood pressure (BP) of >180 mmHg or diastolic BP of >110 mmHg) on the first day of the screening period and on the first day of the treatment period
- (9) Patients for whom any of the following apply upon fundoscopy during the screening period:
  - ✓ No ocular fundus findings are possible.
  - ✓ Active ocular fundus disease
- (10) Patients with severe cardiac failure from the day of consent (Class IV according according to severity classification of the New York Heart Association [NYHA])
- (11) Patients with cerebrovascular disorders or acute coronary syndromes (hospitalization for unstable angina or myocardial infarction, etc.) within 12 weeks prior to the first day of the screening period. Patients who have been hospitalized due to acute coronary angioplasty or cardiac failure.
- (12) Patients with malignant tumors or a history of such. However, this does not apply to patients with no relapse for 5 or more years (5 or more years with no relapse from last administration of chemotherapy if chemotherapy was used).
- (13) Patients with incidence or relapse of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the first day of the screening period
- (14) Patients with current or previous haemosiderosis or hemochromatosis
- (15) Patients with a history of or plans for organ transplant (not including being on a waiting list for renal transplant), haematopoietic stem cell transplant, or bone marrow transplant
- (16) Patients with an allergy to the study drugs
- (17) Patients who have participated in another clinical study and received study drugs within 12 weeks prior to informed consent, or within 5 times the half-life of the study drug (whichever is longer)
- (18) Patients who have previously used MT-6548
- (19) Patients with known low tolerance to HIF-PH inhibitors.
- (20) Patients who are unwilling to consent to use contraception from the beginning of the study period to 30 days following the final dose of the study drug for women who may become pregnant, or from the beginning of the study period to 90 days following the final dose of the study drug for men
- (21) Female patients who are or may be pregnant, or women who are nursing
- (22) Other patients judged by investigators/subinvestigators to be inappropriate as a subject in this study

#### Rationale

- (1)-(4), (6), (18) These were considered likely to affect drug efficacy evaluation of MT-6548.
- (5), (7)–(16), (19) Set in regard for patient safety and ethics.
- (17) Set in regard to ethical performance of study. Also, unevaluated drugs may affect efficacy or safety in unpredictable ways.
- (20) (21) Reproductive and developmental toxicity safety has not been established in humans, and the possibility that the study drug may transfer to human sperm cannot be ruled out. Therefore, this was set for safety reasons.
- (22) Set in order to allow determinations regarding study participation in regard for patient safety for reasons other than the general factors listed above.

#### 3.4 Re-testing/re-screening

#### (1) Re-testing

Re-testing may be performed during the screening period at the discretion of the investigator/subinvestigator for any subject whose laboratory values (Hb, serum ferritin, TSAT, folic acid, vitamin  $B_{12}$ , AST, ALT, and total bilirubin) or BP do not meet the inclusion criteria or meet the exclusion criteria during the screening period.

Subjects with blood pressure measurements on the first day of the treatment period which meet exclusion criteria may be re-tested at the discretion of investigators/subinvestigators, and processed for treatment period initiation if they no longer meet exclusion criteria.

However, the maximum time from the first day of the screening period to the first day of the treatment period is 6 weeks.

#### (2) Re-screening

For any subject whose laboratory values (Hb, serum ferritin, TSAT, folic acid, vitamin B<sub>12</sub>, AST, ALT, and total bilirubin), BP, or BP measurements on the first day of the treatment period do not meet the inclusion criteria or meet the exclusion criteria during the screening period, re-screening may be performed if the investigator/subinvestigator considers that the subject may become eligible for the study due to natural course or with drug therapy.

However, re-screening may only be performed once for any given subject.

#### 4. Explanations to subjects and consent

#### 4.1 Informed consent forms and written information

Study investigators will draft informed consent forms and written information for patients. These will be either a single form, or a set of forms, and will be revised as required.

Authored or revised consent forms will be submitted to study sponsor and approved by the Institutional Review Board (IRB) prior to study initiation.

#### 4.2 Content of written information

Written information for subjects must contain at least the following items:

- (1) The study is for research purposes.
- (2) Study objectives
- (3) Names, titles, and addresses of investigators and subinvestigators
- (4) Study methodology (trial aspects, subject inclusion criteria, and probabilities of being assigned to different study groups).
- (5) Expected clinical benefits, risks, and inconveniences (subjects must also be informed if there are no expected benefits for them)
- (6) If enrolling a patient into the trial, explanation of other therapeutic options for the patient and expected risks/rewards associated with these
- (7) Expected period of study participation for the subject.
- (8) Participation in the study is purely voluntary, and the subject or his/her agent may rescind agreement to participate at any time. If the subject determines not to participate in the study or withdraws consent, he/she will not be disadvantaged in anyway, and will not forego any benefits from not participating.
- (9) Study monitors, auditors, IRB members, and regulatory authorities may view source documents from the study. In this event, subject confidentiality will be preserved. The subject or his/her agent consents to this viewing of source documents by signing (or printing name and affixing personal seal) the consent form.
- (10) Subject confidentiality will be preserved even if study results are published.
- (11) Contact information for consultations with the study center for when subjects wish to learn more information about the study or their rights, or for when study-related damage to health occurs
- (12) Financial reimbursements or treatments available to subjects in the event of damage to health resulting from the study
- (13) Types of IRBs that will investigate and determine issues related to appropriate performance of the study, types of issues which fall under IRB purview, and other study-related issues concerning the IRB
- (14) Planned number of subjects in the study
- (15) If any information comes to light which may affect the willingness of the subject or his/her agent to continue study participation, that information will be rapidly shared with the subject or his/her agent.
- (16) Conditions and reasons leading to study withdrawal
- (17) Details of any costs to be borne by the subject, if applicable
- (18) Details of any money to be paid to the subject, if applicable (agreements for determining amounts, etc.)
- (19) Behaviors or rules to be followed by the subject
- (20) Other necessary items or information related to the study

# 4.3 Method of obtaining consent

- (1) Prior to initiating study, the investigator/subinvestigator will hand the informed consent forms and written information approved by the IRB to each patient in person, and conduct a full explanation. Clinical coordinators may also perform supplementary explanations. Explanations will be based on written information for the study and use as simple language as possible to ensure patient understanding. All patient questions will be answered fully. After confirming that the patient understands fully, he/she may freely grant informed consent for participation in the study in writing.
- (2) The informed consent form will be signed (or names printed and personal seals affixed) and dated by both the patient and the investigator/subinvestigator who performed the explanation. If clinical coordinators performed supplementary explanations, he/she will also sign (or print name and affix personal seal) and date the form.
- (3) If the patient is incapable of reading the written information, the investigator/subinvestigator will arrange for a fair witness to be present when performing the explanation and obtaining consent. In this case, the witness will also sign (or print name and affix personal seal) and date the consent form.
- (4) Before each subject begins participation in the study, the investigator/subinvestigator will issue hand him or her a signed (or names printed and personal seals affixed) and dated copy of the informed consent forms and written information. Originals of the consent forms will be stored at each study center in accordance with that center's regulations.
- (5) The date of informed consent will be recorded on each CRF.

## 4.4 Revision of informed consent forms and written information

- (1) If new significant information is obtained which may impact a subject's consent, investigators/subinvestigators will verbally convey this information to each subject participating in the study in a timely manner, confirm whether the subject wishes to continue participation, and record these actions in the medical records.
- (2) In this event, investigators will determine in a timely manner whether this new information requires revision of informed consent forms and written information.
- (3) If it is determined that informed consent forms and written information must be revised, investigators must make said revisions in a timely manner and obtain approval from the IRB.
- (4) The investigator/subinvestigator must explain relevant information to subjects already participating in the study using revised informed consent forms and written information newly approved by the IRB, and obtain freely-given consent in writing.
- (5) As with the initial informed consent, the revised informed consent form will be signed (or names printed and personal seals affixed) and dated by both the subject and the investigator/subinvestigator who performed the explanation. If clinical coordinators performed supplementary explanations, he/she will also sign (or print name and affix personal seal) and date the form.
- (6) As with the initial informed consent, if the subject is incapable of reading the written information, the investigator/subinvestigator will arrange for a fair witness to be present when performing the explanation and obtaining consent. In this case, the witness will also sign (or print name and affix personal seal) and date the consent form.
- (7) Investigators/subinvestigators will give subjects a signed (or names printed and personal seals affixed) and dated copy of the informed consent forms and written information.
  Originals of the consent forms will be stored at each study center in accordance with that center's regulations.

# 5. Study Design

# 5.1 Study phase and type

Study phase: Phase 3

Study type: Confirmatory study

# 5.2 Study design

This is a multicenter, uncontrolled, open-label study.



#### (1) Screening period

The screening period begins on the first day of the screening period, and ends upon completion of tests required on the first day of the treatment period. Maximum screening period time is 6 weeks. Two visits will be made during the screening period; the first (SV1) is the first day of the screening period. The second screening period visit (SV2) occurs after results from laboratory tests performed on the first day of the screening period have been obtained. Testing may be repeated as necessary.

## (2) Treatment period

The treatment period will last from completion of scheduled tests on the first day of the treatment period to completion of blood sampling for haematology tests on the final day of the treatment period (Week 24 of the treatment period or discontinuation of treatment).

During the treatment period, subjects are to visit the study site on the day of dialysis after a 2-day interdialytic interval; however, if this is difficult, subjects are to visit the study site on the day of dialysis after a 1-day interdialytic interval. After the first day of the treatment period, subjects are to visit the study site every 2 weeks until Week 12 and every 4 weeks after Week 12 to undergo the scheduled test. However, subjects are to visit the study site at shorter intervals as necessary, if excessive increases or decreases in Hb are of concern based on the time course of Hb levels or for hemodialysis.

#### (3) Follow-up observation period

The follow-up observation period consists of 2 weeks from completion of blood sampling for haematology tests on the final day of the treatment period. The final day of the follow-up observation period is 2 weeks from the completion of blood sampling for haematology tests on the final day of the treatment period, regardless of whether a study visit is made on that day.

Subjects should make study visits as close to the same time as possible during the study period for scheduled tests.

#### Rationale

Screening period: Established to confirm subject suitability for the study.

Treatment period: An uncontrolled study design was selected in consideration of feasibility due to the extremely small number of HD-CKD patients in Japan who are not treated with any ESA formulation.

Follow-up observation period: The follow-up observation period for MT-6548 Tablet was set at 2 weeks considering the elimination half-life of MT-6548 in order to investigate AEs occurring after completion of treatment.

# 5.3 Endpoints

## 5.3.1 Efficacy endpoint

- (1) Primary endpoint
  - 1) Mean Hb at treatment period Weeks 20 and 24
  - 2) Hb at each treatment period timepoint
  - 3) Proportion of subjects with mean Hb levels within the target range (10.0–12.0 g/dL), <10.0 g/dL, and  $\ge$ 12.0 g/dL at each timepoint in the treatment period
  - 4) Number of days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL)
  - 5) Rate of increase in Hb levels

#### (2) Other endpoints

- 1) Changes in mean Hb from baseline at treatment period Weeks 20 and 24
- 2) Proportion of subjects with a≥1.0 g/dL increase from baseline in mean Hb levels
- 3) Ratio of subjects who received ESA rescue therapy
- 4) Ratio of subjects who received red blood cell (RBC) transfusion rescue therapy.
- 5) Study drug dosage
- 6) Total number of study drug dosage adjustments

- 7) Quantity of iron administered
- 8) Ratio of subjects with serum ferritin of ≥100 ng/mL or TSAT ≥20%.
- 9) Change from baseline of iron-related measures (serum iron, TIBC, TSAT, and serum ferritin) and hepcidin.
- 10) Change from baseline of haematocrit, RBC count, reticulocytes (counts and fractions), and EPO.
- 11) QOL measures (EQ-5D-5L, KDQOL)

#### Rationale

(1) Primary endpoint

Hb level was set as the primary endpoint because this is already established as the standard assessment measure for nephrogenic anaemia treatment.

(2) Other endpoints

Other endpoints were set in order to enable multifaceted evaluation of changes in Hb, iron-related measures, RBC-related parameters, QOL measures, and concomitant therapies.

## 5.3.2 Safety endpoints

- (1) Adverse events and adverse drug reactions
- (2) Laboratory test values
- (3) Resting standard 12-lead ECG
- (4) Dry weight
- (5) Body weight
- (6) Vital signs
- (7) Fundoscopy
- (8) Chest X-ray
- (9) Proportion of subjects with documented Hb levels of ≥12.0 or ≥13.0 g/dL
- (10) Ratio of subjects with Hb increase rates exceeding 0.5 g/dL/week.

#### Rationale

- (1)–(6) (8) Set to evaluate general safety for HD-CKD patients.
- (7) Set to evaluate effects of MT-6548 on fundus oculi.
- (9) (10) Set to evaluate excessive or acute increase of Hb levels.

# 6. Target sample size and study period

# 6.1 Target sample size

The number of subjects registered in the treatment period will be 20.

## Rationale

The proportion of patients who are not treated with any ESA formulation is as small as approximately 10% of all hemodialysis-dependent patients in Japan. Patients receiving any ESA formulation are allowed to register after undergoing a washout; however, the number of eligible patients was thought to be very limited when considering the selection/exclution criteria. Therefore, the target sample size was set to 20 after consideration of feasibility.

# 6.2 Study period

# 7. Study drug

# 7.1 Study drug names

(1) Investigational product

Name: MT-6548 Tablet 150 mg Nonproprietary name: vadadustat

Dosage form and content: Each film-coated tablet contains 150 mg vadadustat.

# 7.2 Study drug packaging and labelling

(1) Packaging

Each bottle contains 100 tablets of MT-6548.

(2) Labelling

Clinical Study Drugs MT-6548 Tablet 150 mg 100 tablets

Study no.: MT-6548-J04

Lot no.: XXXXX

Storage method: Please store at 1-30°C.

Dosage and administration: Please follow your doctor's instructions.

\*Please return empty bottles and unused study drug.

\*Those not participating in the MT-6548 study must not take the study drugs.

Mitsubishi Tanabe Pharma Corporation, 3-2-10 Dosho-machi, Chuo-ku, Osaka

# 7.3 Storage method

Store between 1-30°C.

# 7.4 Study drug handling, storage, and management methods

The study sponsor will supply study drugs to each study center after conclusion of the study agreement. Study drug managers will follow the Procedures for Management of Study Drug provided by the study sponsor in storage and management of the study drugs, then return all unused study drugs to the monitor.

Investigators/subinvestigators and study drug managers will notify the study sponsor immediately if any abnormalities in study drug quality are discovered. Any such study drug will be returned to the study sponsor as necessary in accordance with the Procedures for Management of Study Drug.

Study drugs must not be used for any other purpose than those described in this protocol (other clinical studies, animal experiments, basic research experiments, etc.).

# 8. Subject-related test methods

# 8.1 Lists of screened subjects, enrolled subjects, and identification codes

The investigator will prepare a list of all patients who received an explanation of the study. All subjects on this list who have granted consent will be assigned an identification code, and a subject identification code list prepared. Key information for comparisons with source documents will be included.

The investigator will also prepare a list of enrolled subjects (including those who withdrew or dropped out), including sex, date of consent, subject identification code, and other information.

# 8.2 Subject enrollment

### 8.2.1 Consent processing and enrollment

- (1) Investigators/subinvestigators will determine which patients are eligible for participation in the study, and obtain written consent as described in "4. Explanations to Subjects and Consent."
- (2) Investigators/subinvestigators will notify the sponsor by fax.
- (3) Patients using ESA formulations will discontinue use and undergo a washout of the designated length.

## 8.2.2 Screening period

(1) Investigators/subinvestigators will confirm patient suitability by the first day of the screening period, determine whether to enroll that patient for the screening period, and notify the sponsor by fax.

\*Notification by fax is not required for re-screening.

## 8.2.3 Treatment period enrollment

- (1) Investigators/subinvestigators will review all laboratory tests and other tests performed up to the first day of the treatment period, and make a suitability determination prior to initiating the treatment period.
- (2) Investigators/subinvestigators will notify the sponsor by fax on the first day of the treatment period.
- (3) Investigators/subinvestigators will take the following actions with the patient depending on the final suitability result.
  - ✓ If determined to be "suitable" to start the treatment period: Transition to the treatment period.

✓ If determined to be "unsuitable" to start the treatment period: Inform patient that they did not meet inclusion criteria and withdraw that patient from the study.

## 8.2.4 Withdrawal processing

(1) Investigators/subinvestigators will notify the sponsor by fax when a patient is withdrawn from the study after informed consent.

# 8.3 Dosage and administration

(1) Initial dose
Single daily dose of 300 mg (2 tablets)

(2) Maintenance dosage and dosage adjustments Maintenance dosage is 150–600 mg once daily and adjusted according to the dosage adjustment guideline below.

## [MT-6548 Tablet dosage adjustment guidelines]

Investigators/subinvestigators will monitor Hb levels throughout the treatment period, and determine whether to adjust study drug dosage or discontinue administration as required. In principle, dosage adjustments should be performed at scheduled visits; however, an unscheduled visit may be provided for dosage adjustment, if considered necessary, in cases where excessive increases or decreases in Hb levels are of concern based on the Hb time course.

Hb levels will be measured in samples collected in the supine position using a HemoCue<sup>®</sup> Hb201 DM analyzer; and in principle, these measurements will be used to determine dosage adjustments. Hb levels on the day of dialysis will be measured in samples collected before dialysis. Hb measurements used for dosage adjustment determinations will be recorded in the subject's CRF. Measurement results from the HemoCue<sup>®</sup> Hb201 DM will be used solely for determination of study drug dosage adjustments, and will not be used for efficacy or safety analysis.

The dosage adjustment algorithm below will be followed in order to improve and maintain Hb levels of 10.0–12.0 g/dL during the study. Dosage steps are defined in the dosage adjustment table below.

MT-6548 Tablet dosage adjustment table

| Step | No. of tablets | Dosage |
|------|----------------|--------|
| 1 | 1 | 150 mg |
| 2 | 2 | 300 mg |
| 3 | 3 | 450 mg |
| 4 | 4 | 600 mg |

\*It is permitted for dosage adjustments not to comply with the dosage adjustment algorithm for safety reasons depending on factors such as clinical status (e.g., AEs, volume depletion, or volume overload), Hb elevation rate, decrease rate, or fluctuations. In such cases, clinical status will be recorded in CRFs. All dosage increases of MT-6548 will be in increments of 1 tablet at a time.

If a dosage increase or reduction according to the dosage adjustment algorithm is impossible because the maximum or minimum dosage on the dosage adjustment table is already being administered, it is permitted to not alter the dosage at that point. However, in this case it will be confirmed whether withdrawal criteria are met, and treatment discontinued if so.

#### MT-6548 Tablet dosage adjustment algorithm

- ✓ Dosage increases should be performed at intervals of at least 4 weeks in principle, and dosage decreases at intervals of at least 2 weeks.
- ✓ If Hb levels suddenly increase (>2.0 g/dL change in the past 4 weeks\*), decrease MT-6548 dosage by 1 tablet.
- ✓ The MT-6548 Tablet dose should be increased by 1 tablet if Hb levels are <10.0 g/dL. However, decrease by 1 tablet instead of increasing in cases of sudden increase in Hb (more than 2.0 g/dL change in past 4 weeks\*).
- ✓ The MT-6548 Tablet dose should be decreased by 1 tablet if Hb levels are >11.5 g/dL.
- ✓ If Hb levels are >12.0 g/dL and ≤13.0 g/dL with a rapid increase in Hb levels (>2.0 g/dL change in the past 4 weeks\*), MT-6548 tablet administration should be discontinued, and the dose should be decreased by 1 tablet and MT-6548 tablet administration resumed after Hb levels decrease to ≤12.0 g/dL.
- ✓ If Hb levels are >13.0 g/dL, MT-6548 tablet administration should be discontinued, and the dose should be decreased by 1 tablet and MT-6548 tablet administration resumed after Hb levels decrease to ≤12.0 g/dL.

\*The rate of increase in Hb levels will be calculated using the Hb levels at the time points closest to 4 weeks among those measured 3–5 weeks prior to the day of dosage adjustment. A rate of change greater than 0.5 g/dL/week will be regarded as a rapid increase in Hb levels. If no Hb levels were measured 3–5 weeks prior to the day of dosage adjustment,

the Hb levels measured at most recent time points prior to 5 weeks before the day of dosage adjustment will be used to calculate the rate of increase in Hb levels.

## (3) Administration method

The study drug is taken once-daily orally. The drug does not need to be taken with meals, but timing should be as consistent as possible throughout the treatment period, both in relation to meals and time of day. (The first dose will be taken after required tests are finished on the first day of the treatment period.)



The dosage adjustment algorithm was set in order to avoid excessive Hb increase with reference to target Hb values in nephrogenic anaemia therapy according to JSDT's "Guideline for Renal Anemia in Chronic Kidney Disease 2015."

# 8.4 Treatment period

From the first day of the treatment period to the day before Week 24 of the treatment period

# 8.5 Concomitant medications and therapies and rescue therapy

## 8.5.1 Prohibited concomitant medications and therapies

#### (1) ESA formulations

Use of ESA formulations will be restricted during the following periods. These restrictions do not apply to rescue therapy.

- 1) Epoetin alpha (recombinant), epoetin beta (recombinant), and epoetin kappa (recombinant): from 1 week prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.
- 2) Darbepoetin alfa (recombinant): from 2 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.
- 3) Epoetin beta pegol (recombinant): from 4 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.

#### (2) Testosterone enanthate and mepitiostane

Concomitant use is prohibited from 8 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period.

## (3) Blood transfusion

Prohibited from 8 weeks prior to the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. These restrictions do not apply to rescue therapy.

## Rationale

(1)–(3) Medications and therapies considered likely to affect evaluation of MT-6548 efficacy are prohibited for concomitant use.

#### 8.5.2 Restricted concomitant medications and therapies

## (1) Iron supplements

From the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period, administer iron supplements to maintain serum ferritin values of  $\geq 100$  ng/mL or TSAT of  $\geq 20\%$ . Iron supplements may be omitted for subjects who respond poorly to them, such as those with an allergy or those with adverse drug reaction (ADRs) to iron (vomiting, etc.).

Investigators/subinvestigators will determine iron supplement dosage and administration route.

Important: Oral iron supplements may impair MT-6548 bioavailability, so oral iron supplements must not be taken at the same time as MT-6548 Tablet. Subjects taking oral iron supplements will be instructed not to take any within 2 hours before or after taking MT-6548 Tablet.

## (2) Iron-containing phosphate binders (ferric citrate hydrate, sucroferric oxyhydroxide)

New use of iron-containing phosphate binders is fundamentally prohibited from the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. If iron-containing phosphate binders are used by a subject on the first day of the screening period, then the same dosage of the same type should fundamentally be continued from the first day of the screening period to completion of blood sampling for haematology tests on the final day of the treatment period. If investigators/subinvestigators determine that a dosage increase is required for iron-containing phosphate binders, then additional treatment will be performed with hyperphosphatemia drugs containing no iron, or treatment switched to hyperphosphatemia drugs containing no iron. Dosage of iron-containing phosphate binders may also be reduced if determined necessary according to the subject's condition. Switching to another hyperphosphatemia drug containing no iron will not be permitted during the period from the first day of the screening period to completion of designated tests for treatment period Week 4.

Important: As with oral iron supplements, iron-containing phosphate binders may impair MT-6548 bioavailability, so iron-containing phosphate binders must not be taken at the same time as MT-6548 Tablet. Subjects taking iron-containing phosphate binders will be instructed not to take any within 2 hours before or after taking MT-6548 Tablet.

## (3) Hemodialysis

The type of hemodialysis is either hemodialysis or hemodiafiltration with a frequency of

three times a week. In principle, a change in the type and frequency of hemodialysis is prohibited from the first day of the screening period to the completion of blood sampling for hematology tests on the final day of the treatment period; however, the type (hemodialysis and hemodiafiltration) and frequency may be changed if the investigator/subinvestigator considers it clinically necessary.

#### Rationale

- (1) Set with reference to criteria for initiating iron supplementation therapy in JSDT's "Guideline for Renal Anemia in Chronic Kidney Disease 2015."
- (2) Continuation of therapy without changing dosage will avoid affecting evaluation of MT-6548 efficacy.
- (3) It was determined that subjects should continue the same type of hemodialysis at the same frequency due to potential effects of changes in these items on evaluation of MT-6548 efficacy.

## 8.5.3 Rescue therapy

The following rescue therapy options will be provided as needed for subject safety. Even if rescue therapies are performed, the subject can continue in the study unless investigators/subinvestigators determine study withdrawal is appropriate. Details of any rescue therapy implemented will be recorded in the subject's CRF.

## (1) ESA formulations

If a subject has received maximum dosages of MT-6548 Tablets for ≥2 weeks and meets all criteria below, the investigator/subinvestigator may administer an ESA as a rescue therapy to improve Hb levels if necessary in order to secure subject safety. An ESA-based rescue therapy may also be provided without meeting the criteria below if the investigator/subinvestigator considers it necessary to secure subject safety, such as in cases of acute decreases in Hb levels. Administration of MT-6548 Tablets will be discontinued when an ESA-based rescue therapy is provided. Administration of MT-6548 Tablets may be resumed after an improvement in Hb levels and should not be coadministered with a rescue therapy with an ESA. Subjects who are not expected to resume administration of MT-6548 Tablets will be withdrawn from the study.

- ✓ Anaemia or anaemia symptoms (e.g., fatigue, weakness, shortness of breath, chest pain, confusion, dizziness) become aggravated compared to the first day of the treatment period to the point they are clinically problematic.
- ✓ Hb levels drop to <8.0 g/dL.
  </p>

#### (2) RBC transfusion

Usually, RBC transfusions are performed when clinically necessary in instances of acute or major bleeding. For less sever anemia, which may be exacerbated, or moderate to severe anemia symptoms, RBC transfusions may be performed as needed clinically at the discretion of the investigator/subinvestigator.

#### (3) Phlebotomy

Phlebotomy may be performed at investigator/subinvestigator discretion in cases of hyperviscosity syndrome, if the rate of Hb increase is concerning to investigators/subinvestigators, or if Hb levels are high enough to warrant concern to investigators/subinvestigators.

#### Rationale

Set out of consideration for subject safety.

## 8.5.4 Recording of concomitant drugs and therapies

The following information will be recorded regarding all concomitant drugs and therapies performed from the first day of the treatment period to completion of the follow-up observation period in the subject's CRF.

Information for the screening period will also be recorded in CRFs regarding drugs described in "8.5.2 Restricted concomitant medications and therapies."

The only information recorded about dialysis, drugs commonly used for dialysis (e.g., dialysate, anticoagulants, and substitution fluid), and physiological saline used for dissolving injectable formulations will be that specified in "9.2.1 Subject background".

- (1) Concomitant drugs: Drug name, daily dosage, administration route, duration of administration, purpose
- (2) Concomitant therapies: Name of therapy, duration of treatment, purpose

# 8.6 Subject oversight

Investigators/subinvestigators, clinical coordinators, or study drug managers will oversee subjects with attention to the following points. Investigators/subinvestigators or clinical coordinators will question subjects about their adherence to the items below.

#### 8.6.1 Drug use guidance for MT-6548 Tablet

Investigators/subinvestigators or study drug managers will give guidance to subjects covering the

following items.

- (1) MT-6548 Tablets will be issued to subjects in bottles containing 100 tablets. If multiple bottles are issued at a time, subjects will open new bottles only after finishing the MT-6548 from the existing bottle. Subjects will bring all bottles of MT-6548 to each study visit for study drug control purposes, including unused bottles, bottles being used, and empty bottles.
- (2) MT-6548 Tablets are to be taken with water once-daily, without chewing. The drug does not need to be taken with meals, but timing should be as consistent as possible throughout the treatment period, both in relation to meals and time of day. If a subject forgets to take the study drug on a given day, they should resume taking the study drug as normal on the next day.
- (3) Oral iron supplements and iron-containing phosphate binders may impair MT-6548 bioavailability, so these must not be taken at the same time as MT-6548 Tablet. Subjects taking oral iron supplements or iron-containing phosphate binders will not take any within 2 hours before or after taking MT-6548 Tablet.

#### 8.6.2 Visits

Subjects should make study visits as close to the same time as possible during the study period for scheduled tests.

## 8.6.3 Lifestyle guidance

Investigators/subinvestigators or clinical coordinators will give guidance to subjects covering the following points.

- (1) Subjects receive examinations and tests on scheduled days. Subjects should always contact the study center if unable to make a scheduled study visit, and follow instructions.
- (2) Subjects should contact investigators/subinvestigators in a timely manner if they experience abnormal symptoms.
- (3) Subjects will receive a study participation card to show when receiving care at other departments or hospitals. Subjects should always inform investigators/subinvestigators or clinical coordinators if they are using any drugs prescribed by other doctors or purchased at a pharmacy. Subjects should always consult with investigators/subinvestigators or clinical coordinators before using any new drugs during the study.
- (4) Maintain the same lifestyle (daily activities, food, etc.) as before to the extent possible.
- (5) Investigators/subinvestigators or clinical coordinators will instruct women who may become pregnant to use the contraception methods described below during the study period and up to 30 days following the final dose of the study drug, and men during the study period and up to

90 days following the final dose of the study drug. Calendar, anovulation, ovulation detection through body temperature, post-ovulation, and withdrawal do not constitute appropriate forms of contraception. This does not apply to postmenopausal women with absence of menstruation for more than 1 year, women with surgical hysterectomy, or women with bilateral ovariectomy.

- 1) Abstain from intercourse
- 2) Use two effective types of contraception. Joint use of a barrier method (latex condoms for men or diaphragm) in conjunction with a highly effective method such as oral contraceptives, IUD, tubal ligation, or vasectomy is recommended.

9. Tests and observations

9.1 Test and observation schedule

| | | Constitute | noring [n] | | | | | 7 | Treatment neriod [h] | ind [h] | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /\text{\rmsign} | Informed | Silliaarse | Screening period [a] | | | ľ | | | atment per | fal nor | | | | | Final day of |
| Item | consent | First day | Visit 2 | First day<br>[b] | W2 | W4 | W6 | W8 | W10 | W12 | W16 | W20 | W24 | Day of<br>discontinuation | the follow-up<br>observation [c] |
| Visit number | IC | IAS | SV2 | IVI | TV2 | TV3 | TV4 | TVS | TV6 | TV7 | TV8 | TV9 | TV10 | TV11 | FU |
| Permitted range (days) | - | - | ٠ | - | #3 | #3 | ±3 | ±3 | #3 | ±3 | 7= | +7 | #7 | +7 or +14 [e] | +7 |
| Procedure/evaluation | | | | | | | | | | | | | | | |
| Informed consent | х | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | х | х | Х | Х | | | | | | | | | | | |
| Patient backgroud and history | х | | | х | | | | | | | | | | | |
| Height | | | | х | | | | | | | | | | | |
| Dry weight, body weight [f] | | | | х | | | | | | x | | | х | Х | |
| Folic acid and vitamin B <sub>12</sub> [g] | | х | | | | | | | | | | | | | |
| Pregnancy tests [i] | | x | | | | | | | | | | | × | Х | |
| Hematology tests [g], [h], [j] | | х | X [k] | х | x | x | × | × | × | × | × | × | × | × | |
| Blood biochemistry tests [g], [h], [l] | | Х | | х | × | х | х | х | х | х | × | x | х | Х | |
| C-reactive protein [g], [h] | | х | | х | | | | | | | | | × | X | |
| Jon-related measures [g], [h] | | Х | | x | × | × | × | × | × | × | × | × | × | × | |
| Hepcidin [h] | | | | x | × | × | × | | | × | | | × | × | |
| EPO [h] | | | | × | × | × | × | | | × | | | × | × | |
| VEGF[h] | | | | × | | | | | | × | | | × | × | |
| Vital signs [g], [h], [m] | | х | | х | х | х | х | x | x | x | × | × | × | X | |
| Resting standard 12-lead ECG[h], [n] | | | | х | | | | | | | | | × | Х | |
| Fundoscopy [e] | | 7 | X | | | | | | | | | X | | X | |
| Chest X-ray [e] | | | x | | | | | | | | | X | | X | |
| Duration of hemodialysis | | | | х | | | | | | | | | × | × | |
| QOL measures (EQ-5D-5L, KDQOL) | | | | × | | | | | | × | | | × | × | |
| AE investigation | | | | × | × | × | × | × | × | × | × | × | × | × | × |
| Blood sampling for genetic analysis [o] | | | | | Blooc | Blood sampling for genetic analysis performed once as early | or genetic a | nalysis per. | formed onc | e as early a | as possible after Week 2 of treatment period | fter Week | 2 of treatm | ent period | |
| Product evaluation/procedure | | | | | | | | | | | | | | | |
| Investigation of concomitant medications/therapies | | | | × | × | × | х | × | × | × | × | × | × | × | × |
| MT-6548 tablets [p], [q] | | | | | | | Administer | ed accordin | g to the do | Administered according to the dosage adjustment guidelines | nent guideli | nes | | | |
| Iron supplements | | | | Iron sup | plements a | Iron supplements administered to maintain serum ferritin values of 2100 ng/mL or TSAT of 220% | to maintair | n serum fer | itin values | of≥100 ng | mL or TSA | \T of ≥20% | ,, | | |

- [a] Maximum screening period length is 6 weeks. Test results will be reviewed prior to transitioning from the first day of the screening period to screening period Visit 2, and from screening period Visit 2 to the first day of the treatment period. Re-testing will be performed as necessary.
- [b] During the treatment period, subjects are to visit the study site on the day of dialysis after a 2-day interdialytic interval; however, if this is difficult, subjects are to visit the study site on the day of dialysis after a 1-day interdialytic interval.
- [c] Not required if withdrawn prior to the treatment period.
- [d] To be perform prior to the study drug treatment (AE investigation begins after study drug administration).
- [e] Fundoscopy and chest X-ray performed once during screening period, once during Weeks 20–24 of treatment period. In the case of discontinuation of the treatment period, fundoscopy and chest X-ray should be performed within 14 days after discontinuation whenever possible.
- [f] Body weights should be measured before and after dialysis.
- [g] To be measured before dialysis on the day of dialysis during the screening period.
- [h] Tests during the treatment period should be performed before dialysis on the day of dialysis.
- [i] To be performed only in female subjects of childbearing potential.
- [i] Hb levels should be measured in blood collected in the supine position.
- [k] Only Hb levels should be measured.
- [1] Only urea nitrogen levels should be measured before and after dialysis on the first day, Week 24 of the treatment period, and on the day of treatment discontinuation.
- [m] To be measured in the sitting position after a 5-minute rest before blood sampling whenever possible.
- [n] To be measured in the supine position after a 5-minute rest before blood sampling whenever possible.
- [o] For subjects giving consent to blood sampling for genetic analysis, blood will be collected once as early as possible after Week 2 of the treatment period.
- [p] MT-6548 Tablets should be prescribed depending on the number of unused tablets by the subject. Subjects should be instructed to open a new bottle after using up the tablets in one bottle.
- [q] In principle, dosage adjustments should be performed at scheduled visits; however, an unscheduled visit may be provided for dosage adjustment, if considered necessary, in cases where excessive increases or decreases in Hb levels are of concern based on the Hb time course.

If tests and observations cannot be performed on the scheduled day, they may be performed within the permitted ranges shown below. During the treatment period, subjects are to visit the study site on the day of dialysis after a 2-day interdialytic interval; however, if this is difficult, subjects are to visit the study site on the day of dialysis after a 1-day interdialytic interval.

Table 9.1-1 Permitted ranges for study center visits

| Evalu | ation timepoint | Reference date | Permitted range |
|---|---|---|---|
| Screening | First day | | _ |
| period* <sup>1</sup> | Visit 2 | _ | _ |
| | First day*2 | Day 0 | <del>-</del> |
| | Week 2 | Day 14 | Day 11–17 |
| | Week 4 | Day 28 | Day 25–31 |
| | Week 6 | Day 42 | Day 39–45 |
| Transfers out a suis d | Week 8 | Day 56 | Day 53–59 |
| Treatment period | Week 10 | Day 70 | Day 67–73 |
| | Week 12 | Day 84 | Day 81–87 |
| | Week 16 | Day 112 | Day 105–119 |
| | Week 20 | Day 140 | Day 133–147 |
| | Week 24 | Day 168 | Day 161–175 |
| Day of discontinuation of treatment | | Day of | Within 7 days of |
| | | discontinuation | discontinuation*3 |
| | | Week 24 of | |
| Follow-up | | treatment period | |
| observation | Day of completion | (or day of | 14–21 days |
| period | | discontinuation of | |
| | | treatment period) | |

<sup>\*1:</sup> Maximum screening period length is 6 weeks. Re-testing may be performed as necessary.

<sup>\*2:</sup> The first day of the treatment period is defined as the day the investigator/subinvestigator determined the subject to be "suitable" to start the treatment period.

<sup>\*3:</sup> Fundoscopy and chest X-ray to be performed to extent possible within 14 days of study withdrawal.

# 9.2 Test and observation timepoints

## 9.2.1 Subject background

The following subject background factors will be determined and recorded in the CRF.

- (1) Sex
- (2) Date of birth (western calendar)
- (3) Height
- (4) Race
- (5) Ethnicity
- (6) Smoking status
- (7) Underlying cause of CKD
- (8) Time of onset of nephrogenic anaemia
- (9) Concomitant illnesses (illnesses present on the first day of the treatment period)
- (10) Start time of hemodialysis
- (11) Type of hemodialysis\* (hemodialysis or hemodiafiltration)
- (12) Frequency of hemodialysis\*2 (times/week)
- (13) Hemodialysis conditions (dialyzer, dialysate, type of anticoagulant)
- (14) ESA formulation washout (yes/no)
- (15) Type, administration route, dose interval, dosage, and final day of ESA formulation washed out
- \*1: If the type of hemodialysis is changed at any point from the first day of the treatment period to the final day of the follow-up observation period, the date of the change and the type after the change should be recorded in the CRF.
- \*2: If the frequency of hemodialysis is changed at any point from the first day of the treatment period to the final day of the follow-up observation period, the date of the change and the frequency after the change should be recorded in the CRF.

#### 9.2.2 Treatment status

The following information should be recorded in CRFs.

- (1) MT-6548 dosage (details and reasons for change if there was a change of dosage or drug holiday)
- (2) First day of MT-6548 treatment and final day of MT-6548 treatment
- (3) MT-6548 treatment compliance status
- (4) Timing of MT-6548 doses (pre-prandial: within 30 minutes prior to eating; post-prandial: within 30 minutes of eating (including eating); other)

#### (5) MT-6548 dose date and time\*

\* Date and time of dose immediately prior to blood sampling for EPO measurement at treatment period Weeks 2, 4, 12, and 24, and day of discontinuation.

## 9.2.3 Efficacy endpoints

Blood sampling will be performed at each study center for measurement by the contract laboratory testing facility. Study centers will store test reports issued by the contract testing laboratory.

During the screening period, blood will be collected before dialysis whenever the subject makes a study visit on the same day they are scheduled for dialysis. During the treatment period, blood will be collected before dialysis on days the subject is scheduled for dialysis.

#### (1) Hb value

Blood sampling and Hb measurement will be performed in the supine position on the first day of the screening period, screening period Visit 2, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment.

## (2) Ratio of subjects who received ESA rescue therapy

If ESA rescue therapy is performed, type of ESA formulation used, administration route, dose interval, and dosage will be recorded in the CRF.

#### (3) Ratio of subjects who received red blood cell (RBC) transfusion rescue therapy.

If RBC transfusion rescue therapy is performed, type of RBC formulation used and dosage will be recorded in the CRF.

## (4) Study drug dosage

Study drug dosage will be recorded in CRFs.

#### (5) Total number of dosage adjustments

Yes/no for study drug dosage adjustments and post-adjustment dosage will be recorded in the CRF.

## (6) Quantity of iron administered

Iron dosage will be recorded in CRFs.

### (7) Iron-related measures (serum iron, TIBC, TSAT, and serum ferritin)

Blood sampling and measurement will be performed for serum iron, TIBC, TSAT, and serum ferritin on the first day of the screening period, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment.

#### (8) Hepcidin

Blood sampling and measurement of hepcidin will be performed on the first day of the treatment period, treatment period Weeks 2, 4, 6, 12, and 24, and the day of discontinuation of treatment.

### (9) Haematocrit, RBC count

Blood sampling and measurement will be performed for haematocrit and RBC count on the first day of the screening period, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment.

#### (10) Reticulocytes (counts and fractions)

Blood sampling and measurement will be performed for reticulocytes (counts and fractions) on the first day of the screening period, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment.

## (11) EPO

Blood sampling and measurement of EPO will be performed on the first day of the treatment period, treatment period Weeks 2, 4, 6, 12, and 24, and the day of discontinuation of treatment. Blood sampling time will be recorded in CRFs.

## (12) QOL measures (EQ-5D-5L, KDQOL)

Subjects will fill out EQ-5D-5L and KDQOL questionnaires (Appendices 4 and 5) on the first day of the treatment period, treatment period Weeks 12 and 24, and the day of discontinuation of treatment, and results recorded in CRFs.

## 9.2.4 Safety endpoints

## 9.2.4.1 Objective findings

#### (1) Laboratory tests

The following laboratory parameters will be measured at a contract testing laboratory following blood collection at the study center. Study centers will store test reports issued by the contract testing laboratory.

During the screening period, blood will be collected before dialysis whenever the subject makes a study visit on the same day they are scheduled for dialysis. During the treatment

period, blood will be collected before dialysis on days the subject is scheduled for dialysis. Only urea nitrogen levels should be measured before and after dialysis on the first day, Week 24 of the treatment period, and on the day of treatment discontinuation.

Investigators/subinvestigators will record day of confirmation and confirmation results (clinical significance) for the following tests.

#### 1) Haematology tests:

Blood sampling and measurement will be performed for the following parameters on the first day of the screening period, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment.

Parameters: Mean corpuscular volume, mean cell haemoglobin, mean cell haemoglobin concentration, red cell distribution width, WBC count, WBC fraction (neutrophils, eosinophils, monocytes, lymphocytes, basophils), platelet count

#### 2) Blood biochemistry tests:

Blood sampling and measurement will be performed for the following parameters on the first day of the screening period, the first day of the treatment period, Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the treatment period, and the day of discontinuation of treatment. Only urea nitrogen levels should be measured before and after dialysis on the first day, Week 24 of the treatment period, and on the day of treatment discontinuation.

Parameters: Total protein, albumin, blood glucose, urea nitrogen, creatinine, uric acid, CPK, total bilirubin, AST, ALT, ALP, LDH, γ-GTP, Na, K, Cl, Ca, P, Mg, bicarbonate, total cholesterol, LDL-C, HDL-C, triglycerides

#### 3) C-reactive protein:

Blood sampling and measurement of C-reactive protein will be performed on the first day of the screening period, the first day of the treatment period, treatment period Week 24, and the day of discontinuation of treatment.

#### 4) Folic acid and vitamin $B_{12}$ :

Blood sampling and measurement of folic acid and vitamin  $B_{12}$  will be performed on the first day of the screening period.

#### 5) Vascular endothelial growth factor (VEGF)

Blood sampling and measurement of VEGF will be performed on the first day of the screening period, treatment period Weeks 12 and 24, and the day of discontinuation of treatment.

#### (2) Resting standard 12-lead ECG

Resting standard 12-lead ECG will be measured in the supine position during hospital visits on the first day of the treatment period, treatment period Week 24, and the day of discontinuation of treatment ECG diagnosis consists of a comprehensive evaluation including arrhythmia and wave-form diagnoses.

Measured to extent possible prior to blood sampling before dialysis on the day of dialysis. Measurements will be made before blood sampling when possible, and after 5 minutes at rest.

- 1) Normal
- 2) Clinically non-problematic abnormality
- 3) Clinically problematic abnormality

## (3) Dry weight

Dry weight will be measured during study visits on the first day of the treatment period, treatment period Weeks 12 and 24, and the day of discontinuation of treatment. Measurements are recorded in CRFs.

#### (4) Body weight

Body weight will be measured before and after dialysis during study visits on the first day of the treatment period, treatment period Weeks 12 and 24, and the day of discontinuation of treatment. Measurements are recorded in CRFs.

## (5) Duration of hemodialysis

The duration of hemodialysis during visits on the first day, Week 24 of the treatment period, and on the day of treatment discontinuation should be recorded in CRFs.

#### (6) Vital signs

Sitting blood pressure and pulse rate will be measured during study visits on the first day of the treatment period, treatment period Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24, and the day of discontinuation of treatment.

During the screening period, measurements will be made before dialysis whenever the subject makes a study visit on the same day they are scheduled for dialysis. During the treatment period, measurements will be made before dialysis on days the subject is scheduled for dialysis. Measurements will be made before blood sampling when possible, and after 5 minutes at rest.

## (7) Fundoscopy

Fundoscopy will be performed once each within the screening period, from treatment period Week 20 to Week 24, and to extent possible within 14 days of study withdrawal. An ophthalmologist will perform the fundoscopy and make evaluations according to the 3-point scale below. Ophthalmologist evaluations will be recorded in CRFs. Fundoscopy images and ophthalmologist evaluations will be stored at study centers.

- 1) Normal
- 2) Clinically non-problematic abnormality
- 3) Clinically problematic abnormality (retinal hemorrhage yes/no, retinal oedema yes/no)

#### (8) Chest X-ray

Fundoscopy will be performed once each within the screening period, from treatment period Week 20 to Week 24, and to extent possible within 14 days of study withdrawal. Investigators/subinvestigators will evaluate test results according to the 3point scale below. Evaluation results will be recorded in CRFs. Chest X-rays will be stored at the study center.

- 1) Normal
- 2) Clinically non-problematic abnormality
- 3) Clinically problematic abnormality

## (9) Pregnancy tests (only for women who may become pregnant)

Blood sampling and pregnancy testing will be performed on the first day of the screening period, treatment period Week 24, and the day of discontinuation of treatment. Investigators/subinvestigators will evaluate pregnancy based on test results and interview when appropriate. Evaluation results will be recorded in CRFs. If the subject is incapable of becoming pregnant, the reason for this will be recorded in CRFs (women only).

#### 9.2.4.2 Adverse events

AEs are all clinically problematic or unplanned signs (including clinically significant abnormal laboratory values), symptoms, or illnesses occurring after administration of the study drug during the safety evaluation period, regardless of causal relationship with the study drug. Instances of aggravation of events (in terms of severity or seriousness) are treated as new AEs.

However, AEs occurring from informed consent to the first day of the treatment period which match criteria for serious adverse events are still reported to the study sponsor according to "11.1 Responses to occurrence of serious adverse events."

## (1) Symptoms and diseases

Investigators/subinvestigators will confirm AEs through interviews and examinations.

#### (2) Objective findings

Objective findings determined clinically problematic abnormalities\* by investigators/subinvestigators are treated as AEs.

\*Clinically problematic abnormalities are determined according to the following criteria.

- If related to clinical signs or symptoms.
   However, if the sign or symptom has already been separately reported as an AE, the relevant laboratory test abnormality does not require treatment as adverse event.
- If the relevant laboratory test abnormality was treated medically or surgically.
- If the relevant laboratory test abnormality causes a change in method of administration of the study drug (dosage change, drug holiday, discontinuation, etc.).
- If investigators/subinvestigators otherwise determine the abnormality to be clinically problematic.

## (3) Adverse event evaluation and standards

1) Date of onset

Date the symptom or laboratory test abnormality was observed.

#### 2) Severity

Adverse event severity is classified as follows:

- 1. Mild: No effect on activities of daily life
- 2. Moderate: Moderate impairment of activities of daily life caused by event
- 3. Severe: Event prevents performing activities of daily life

#### 3) Seriousness

AE seriousness is classified as follows:

- 1. Not serious: Any events other than 2 below.
- 2. Serious: Any events (a) to (f):
- (a) Fatal
- (b) Life-threatening
- (c) Necessitating hospitalization or prolongation of hospitalization for treatment
- (d) Events leading to permanent or clear dysfunction or disability
- (e) Other events or reactions judged medically significant

## (f) Causing congenital anomalies or defects

## 4) Causal relationship with the study drug

The investigator/subinvestigator will assess whether or not there is a logical possibility that the study drug caused the AE. This assessment will take into account factors not related to the study drug, including risk factors such as natural course and concurrent treatments for underlying or concomitant diseases, as well as the temporal relationship between the study drugs and the event (recurrence after resuming administration, elimination after discontinuation, etc.). AEs for which a logical possibility of a causal relationship with the study drug exists will be treated as ADRs.

- 1. Logical possibility
- 2. No logical possibility

#### 5) Outcome

AE outcomes are classified as follows:

- 1. Recovery
- 2. Relief
- 3. Not recovered
- 4. Recovered with sequelae
- 5. Death
- 6. Unknown

#### 6) Date of outcome

Date of outcome is determined according to the following criteria:

Recovery: Date of recovery. If date of recovery is knot known, use date on which recovery was confirmed or determined.

Relief: Date on which relief was confirmed or determined.

Not recovered: Date on which "not recovered" was confirmed or determined.

Recovered with sequelae: Date on which "recovered with sequelae" was confirmed or determined.

Death: Date of death. If date is not known, use date of confirmation or determination.

Unknown: Date of death if outcome is unknown due to death of subject for cause other than the relevant AE. For other circumstances use date of confirmation or determination.

## 7) Action taken with the study drug

Actions taken with the study drug are classified into the following 6 categories:

- 1. Discontinuation of administration (study withdrawal)
- 2. Drug holiday
- 3. Dosage increase
- 4. Dosage reduction
- 5. No action
- 6. Not applicable (occurred after final administration of study drug)

## 8) Actions taken other than with the study drug

Actions taken other than with the study drug are classified into the following two categories: If actions other than with the study drug were taken, details of these will be investigated and recorded in the CRF.

- 1. No
- 2. Yes

## 9) Follow-up investigation



- Period [1] above is the 14 days from the day after completion of the treatment period, during which any AEs will be investigated.
- Period [2] above is the 28 days from the day after completion of the follow-up observation period; it is the period for follow-up investigations of AEs occurring during the safety evaluation period (treatment period + Period [1]).
- Course of AEs subject to follow-up investigation during Period [2] are recorded in the subject's CRF. The date of outcome written in the CRF for AEs with outcomes of relief or not recovered is the day of observation after completion of Period [2], during Period [3].
- Further investigations (Period [3]) will be performed for the course of ADRs with outcomes of relief or not recovered as of the end of Period [2].

- If there is a valid reason to halt investigations mid-way after completion of the safety evaluation period (after completion of Period [1]), record reasons for this and conclude the follow-up investigation.

## (4) Recording information in CRFs

If an AE is observed, investigators/subinvestigators will record the following information in the subjec's CRF: name of AE\*, date of onset, severity, seriousness, causal relationship with study drug, details of any actions taken (drug names, treatment methods, etc.), outcome, and date of outcome.

- \*AE names are handled in the following manner:
- Fundamentally, the name of diagnosis is used.
- The symptom name is used if a clear diagnosis has not been made.
- If there are multiple symptoms which can be expressed by a one diagnosis, that diagnosis name is used
- Medical treatments etc. are not considered AEs; rather the disease or symptom requiring surgical treatment is considered the AE.

## 9.2.5 Blood sampling for genetic analysis

Blood sampling for genetic analysis will be performed once as early as possible after Week 2 of treatment period in subjects who have granted consent to genetic analysis. The blood sampling volume will be about 8.5 mL (refer to "25. Genetic analysis study").

## 10. Evaluation methods and standards

## 10.1 Efficacy

#### 10.1.1 Primary endpoint

The following endpoints will also be studied.

Mean Hb at treatment period Weeks 20 and 24
 Mean Hb of treatment period Weeks 20 and 24 will be calculated.

(2) Hb at each treatment period timepoint

Hb at each timepoint in treatment period will be calculated.

- (3) Proportion of subjects with mean Hb levels within the target range (10.0–12.0 g/dL),
  - <10.0 g/dL, and ≥12.0 g/dL at each timepoint in the treatment period

Ratios of subjects with mean Hb within the target range (10.0–13.0 g/dL), <10.0 g/dL, and >12.0 g/dL at each timepoint in treatment period will be calculated.

(4) Number of days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL)

Number of days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL) will be calculated.

(5) Rate of increase in Hb levels

The rate of increase in Hb levels will be calculated using the following methods.

- ✓ The change in Hb level from the first day of the treatment period to treatment period Week 4 will be calculated.
- ✓ Calculated from the slope of the regression line obtained from Hb levels on the first day of the treatment period and at treatment period Weeks 2, 4, and 6.

## 10.1.2 Other endpoints

The following endpoints will also be studied.

(1) Changes from baseline in mean Hb levels at Weeks 20 and 24 of the treatment period Changes from baseline in mean Hb levels at Weeks 20 and 24 of the treatment period will be calculated. (2) Proportion of subjects with a ≥1.0 g/dL increase from baseline in mean Hb levels at Weeks 20 and 24 of the treatment period

Proportion of subjects with a ≥1.0 g/dL increase from baseline in mean Hb levels at Weeks 20 and 24 of the treatment periodwill be calculated

(3) Ratio of subjects who received ESA rescue therapy

Ratio of subjects who received ESA rescue therapy from the first day of the treatment period to treatment period Week 24 will be calculated.

(4) Ratio of subjects who received red blood cell (RBC) transfusion rescue therapy.

Ratio of subjects who received RBC transfusion from the first day of the treatment period to treatment period Week 24 will be calculated.

(5) Study drug dosage

Mean daily dosage will be calculated for each scheduled study visit from the first day of the treatment period up to treatment period Week 24.

(6) Total number of study drug dosage adjustments

The total number of dosage adjustments from the first day of the treatment period to treatment period Week 24 will be calculated.

(7) Quantity of iron administered

Mean weekly dosage will be calculated for each scheduled study visit from the first day of the treatment period up to treatment period Week 24.

(8) Ratio of subjects with serum ferritin of  $\geq$ 100 ng/mL or TSAT  $\geq$ 20%.

Ratio of subjects with serum ferritin of  $\geq 100$  ng/mL or TSAT  $\geq 20\%$  at each evaluation timepoint will be calculated.

(9) Change from baseline of iron-related measures (serum iron, TIBC, TSAT, and serum ferritin) and hepcidin.

Changes in iron-related measures (serum iron, TIBC, TSAT, and serum ferritin) and hepcidin from baseline will be calculated for each evaluation timepoint.

(10) Change from baseline of haematocrit, RBC count, reticulocytes (counts and fractions), and EPO.

Changes in haematocrit, RBC count, reticulocytes (counts and fractions), and EPO from

baseline will be calculated for each evaluation timepoint.

# (11) QOL measures (EQ-5D-5L, KDQOL)

Scores for QOL measures will be calculated for each evaluation timepoint.

# 10.2 Safety

The following endpoints will also be studied.

- (1) AEs and ADRs (refer to "9.2.4.2 Adverse events" for details)
- (2) Laboratory test values
- (3) Resting standard 12-lead ECG
- (4) Dry weight
- (5) Body weight
- (6) Vital signs
- (7) Fundoscopy
- (8) Chest X-ray
- (9) Proportion of subjects with documented Hb levels of ≥12.0 or ≥13.0 g/dL
- (10) Ratio of subjects with Hb increase rates exceeding 0.5 g/dL/week.

## 11. Ensuring subject safety

# 11.1 Responses to serious adverse events

If an SAE occurs after informed consent is granted, investigators/subinvestigators will immediately take appropriate actions toward the subject regardless of causal relationship with the study drug.

Investigators/subinvestigators will immediately notify monitors once an SAE has occurred (fundamentally in writing), and make a detailed written report to the study sponsor within 7 days of this report. Investigators/subinvestigators will also report the SAE to the director of the applicable study center.

[Definition of serious adverse events]

- (1) Fatal
- (2) Life-threatening
- (3) Necessitating hospitalization or prolongation of hospitalization for treatment
- (4) Events leading to permanent or clear dysfunction or disability
- (5) Other events or reactions judged medically significant
- (6) Causing congenital anomalies or defects

# 11.2 Significant adverse events

There are no SAEs which should be defined with regard to studying the safety profile of the drug.

## 11.3 Pregnancy reporting

If investigators/subinvestigators learn that a female subject or the female partner of a male subject may have exposed an embryo or fetus to the study drug from the first day of the treatment period to the end of the contraception period, they will immediately inform the study sponsor using Pregnancy Reports (Appendix 1). If the female subject or female partner of a male subject wishes to deliver the baby, investigators/subinvestigators will to the extent possible perform follow-up investigation up to birth in order to investigate effects of the study drug on the newborn. Results of the investigation will be reported to the study sponsor using Pregnancy Reports (Appendix 1).

# 11.4 Contacting subjects' other doctors

Investigators/subinvestigators will confirm whether or not each subject is receiving medical care other than as part of the current study during the study period. If a subject is receiving such care, the other doctor will be contacted with the consent of the subject and informed of the subject's

participation in the study. In order to enlist subject aid in contacting other doctors, the investigators/subinvestigators or clinical coordinators may give each subject a card for the current study, and request that the subject show this to other hospitals or departments.

# 12. Withdrawal criteria and procedures

#### 12.1 Withdrawal criteria

Subjects will be withdrawn from the study if the following criteria are met:

- (1) If the subject expresses a desire to withdraw from the study.
- (2) If it is discovered that the subject is clearly ineligible for study participation.
- (3) If investigators/subinvestigators determine that AEs make continued participation in the study difficult.
- (4) If investigators/subinvestigators determine that continuation of the study is inappropriate for a subject, such as if hyperviscosity syndrome occurs or if control of Hb within the target range is impossible.
- (5) If the subject no longer requires hemodialysis or hemodiafiltration.
- (6) If the subject has undergone renal transplantation.
- (7) If pregnancy of the subject is discovered.
- (8) If the investigator/subinvestigator determines a subject should withdraw from the study for any other reason.

#### Rationale

- (1) Set out of ethical considerations.
- (2) (5) (6) Set in order to prevent study drug administration to subjects unsuitable for inclusion in safety or efficacy evaluation.
- (3) (4) (7) Set out of safety considerations.
- (8) Set in order to allow the investigator/subinvestigator to make determinations regarding study continuation for significant safety-related reasons other than those enumerated above.

## 12.2 Procedures for withdrawal

When withdrawing a subject from the study, investigators/subinvestigators will take appropriate measures with that subject, promptly notify the monitor of the reason for withdrawal, and notify the sponsor by fax in accordance with Section "8.2.4 Withdrawal processing." Investigators/subinvestigators will also perform designated tests and observations to be completed within 7 days of withdrawal from the treatment period (funduscopy and chest X-ray should be performed within 14 days of withdrawal from the treatment period whenever possible).

Investigators/subinvestigators will record date of withdrawal and reasons for withdrawal in the CRF for subjects who withdraw from the study following the first day of the treatment period. If the reason for withdrawal is an AE, the name of the event will be recorded in the CRF. The date of evaluations performed upon withdrawal is used as the date of withdrawal, but if these evaluations
could not be performed, the date of determination of withdrawal may be used instead. If tests and observations required on the day of withdrawal cannot be performed for a given subject, or the subject does not make any post-withdrawal visits, follow-up investigation will be performed through correspondence (sealed letters) or telephone to ascertain reasons for this and subsequent course, and information obtained recorded.

#### 13. Statistical analysis

# 13.1 Analysis sets

Efficacy analysis is performed with the full analysis set (FAS). Safety analysis will be performed with the safety analysis set.

The analysis sets are defined as follows. However, details regarding subjects handling will be determined by the sponsor before data lock.

#### (1) FAS

The FAS consists of all subjects who transitioned to the treatment period excluding the following subjects:

- ✓ Subjects who did not have HD-CKD-related anaemia
- ✓ Subjects who did not use a single dose of study drug
- ✓ Subjects with absolutely no efficacy data after start of study drug administration

#### (2) Safety analysis set

The safety analysis set consists of all subjects who transitioned to the treatment period excluding the following subjects:

- ✓ Subjects who did not use a single dose of study drug
- ✓ Subjects with absolutely no safety data after start of study drug administration

#### 13.2 Data handling

#### (1) Definition of missing values

If test measurements are missing or if problems with samples etc. result in invalid measurements or reference values, these are handled as missing values.

#### (2) Handing of timepoint data for statistical summaries at each measurement timepoint

Statistical summaries for each evaluation timepoint will use data compliant with permitted ranges as described in "Table 9.1-1 Permitted ranges for study center visits." There will be no supplementing with data from outside the permitted range.

If multiple data points exist within the permitted range, then the one closes to the scheduled day will be used. If there are deviations from the scheduled day, then data points prior to the scheduled day will be used for efficacy evaluation, and data points after the scheduled day will used for safety evaluation.

#### (3) Handling of efficacy endpoints if rescue therapy was implemented

No data obtained after implementation of rescue therapy will be used for efficacy evaluation.

#### (4) Imputation of missing values

Missing values for treatment period Week 24 will be imputed by last observation carried forward (LOCF). Data from treatment period Week 24 with missing values imputed will be used as data from the completion of treatment period.

Required regulations for data handling other than those enumerated above will be described in the statistical analysis protocol prior to data lock.

# 13.3 Statistical analysis protocol

Confidence interval will be 2-sided, with a confidence coefficient of 95%. Data imputed using LOCF will not be used in analysis with mixed models repeated measures (MMRM).

A detailed statistical analysis protocol will be authored prior to data lock.

#### 13.3.1 Demographic and other baseline characteristics

Summary statistics will be compiled for demographic data and other baseline characteristics for all analysis sets. Incidence and ratios will be shown for discrete data, while descriptive statistics will be calculated for continuous data (number of subjects, mean, SD, minimum, median, maximum, and 95% CI for means, same below).

# 13.3.2 Efficacy

#### (1) Analysis methods for primary endpoint

1) Mean Hb at treatment period Weeks 20 and 24

For mean Hb at treatment period Weeks 20 and 24, mean Hb at each timepoint will be modeled using MMRM with the following model, and mean Hb at treatment period Weeks 20 and 24 and their two-sided 95% CI will be calculated.

#### [MMRM model]

- > Fixed effects: Evaluation timepoint
- > Random effects: Subjects

#### 2) Hb at each treatment period timepoint

Descriptive statistics will be calculated for Hb levels at each treatment period timepoint, and analysis performed taking into account changes over time using MMRM.

- 3) Proportion of subjects with mean Hb levels within the target range (10.0–12.0 g/dL), <10.0 g/dL, and ≥12.0 g/dL at each timepoint in the treatment period Numbers and ratios of subjects with mean Hb at each treatment period timepoint within the target range (10.0–12.0 g/dL), <10.0 g/dL, and ≥12.0 g/dL will be shown.</p>
- 4) Number of days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL)

Descriptive statistics will be calculated for days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL). A Kaplan-Meier plot will be shown for days from the first day of the treatment period required to reach the target Hb range (10.0–12.0 g/dL). Statistical summaries will not include subjects with Hb  $\geq$ 10.0 g/dL on the first day of the treatment period.

5) Rate of increase in Hb levels

Descriptive statistics will be calculated for the rate of increase.

(2) Other endpoints

Incidence and ratios will be shown for discrete data, while descriptive statistics will be calculated for continuous data.

#### 13.3.3 Safety

(1) Analysis methods for AEs and ADRs

The following statistics will be shown: numbers of subjects and incidence ratios for AEs, SAEs, AEs leading to discontinuation, AEs leading to death, ADRs, serious ADRs, ADRs leading to discontinuation, and ADRs leading to death.

(2) Analysis methods for laboratory values, resting standard 12-lead ECG, dry weight, body weight, vital signs, fundoscopy, and chest X-ray

Descriptive statistics will be calculated for continuous data at each timepoint. Descriptive statistics will also be calculated for changes from baseline. A shift table will be shown for changes of discrete data from baseline to each timepoint.

(3) Analysis methods for ratios of subjects with Hb levels of  $\geq$ 12.0 g/dL or  $\geq$ 13.0 g/dL.

Numbers and ratios of subjects with Hb levels of  $\geq$ 12.0 g/dL or  $\geq$ 13.0 g/dL at each timepoint will be shown.

(4) Ratio of subjects with Hb increase rates exceeding 0.5 g/dL/week.

Numbers and ratios of subjects with rate of Hb increase of >0.5 g/dL/week will be shown.

# 13.4 Changes in statistical analysis protocol

If any portion of the statistical analysis plan is modified prior to data lock, reasons for change will be described in the statistical analysis protocol and the clinical study report. If the analysis plan is modified or analyses added after data lock, reasons for modification will be described in the statistical analysis protocol and the clinical study report, and analytical results will be distinguished from the original plan.

# 14. Study protocol compliance, deviation, and modification

# 14.1 Study protocol agreement and compliance

Before each investigator agrees with the study sponsor about the study protocol, he or she will discuss it with the study sponsor based on the protocol, newest investigator's Brochure (IB), and other materials provided. The investigator must fully study the ethical and scientific validity of the study prior to agreement.

In order to demonstrate agreement with the study sponsor on the study protocol and intent to comply with it based on these considerations, the investigator will sign (or print name and affix personal seal) the Agreement and enter the date with the study sponsor.

# 14.2 Study protocol deviations and modifications

Investigators/subinvestigators may not deviate from or modify the study protocol without previous written permission from the study sponsor and IRB. However, if there are circumstances in which such a deviation or modification is medically necessary on an emergency basis to avoid placing subjects in danger, investigators/subinvestigators may perform such actions without prior permission from the study sponsor and IRB.

In such cases, investigators must submit and receive approval for said deviations or modifications, reasons for these, and if appropriate revisions to the study protocol as rapidly as possible from the study sponsor, study center director, and the IRB. Approval from the study center director and agreement from the study sponsor must be obtained in writing.

Investigators/subinvestigators shall fully record all actions deviating from the study protocol.

Investigators shall also draft a report detailing all medically required emergency deviations from or modifications to the study protocol for the purpose of avoiding placing subjects in danger, including the reasons why they were necessary. Investigators will keep a copy of this report and send it to the study sponsor and study center director.

Investigators must immediately submit a report to the study sponsor, study center director, and IRB about all modifications which may significantly influence the study or increase risk to subjects.

# 15. Revisions to the study protocol

The study sponsor may revise the study protocol during the study if modifications are required. The study sponsor will discuss the revisions with investigators and come to agreement about them, then immediately notify the study center director in writing and obtain approval from the IRB through the study center director.

If the study center director requests modification of the protocol based on the opinion of the IRB, the study sponsor will determine whether the modification is warranted and revise the protocol as necessary. The study sponsor will discuss the revisions with investigators and come to agreement about them, then immediately notify the study center director in writing and obtain approval from the IRB through the study center director.

If investigators request modification of the protocol, the study sponsor will determine whether the modification is warranted and revise the protocol as necessary. The study sponsor will discuss the revisions with investigators and come to agreement about them, then immediately notify the study center director in writing and obtain approval from the IRB through the study center director.

# 16. Termination or suspension of the entire study

- (1) Standards for termination or suspension of the study In the following circumstances the study sponsor will determine whether or not continuation of the study is warranted at some or all study centers.
  - 1) If significant information is learned about study drug quality, efficacy, or safety, or if other information about appropriate conduct of the study comes to light.
  - 2) If modifications to the study protocol are required which study centers cannot adopt.
  - 3) If a study center director requests modifications to the study protocol based on the opinion of the IRB, but the study sponsor cannot accept these changes.
  - 4) If a study center director orders termination of the study based on the judgment of the IRB.
  - 5) If a study center makes significant or continued deviations from GCP, the current study protocol, or the study contract.

#### (2) Termination or suspension of the entire study by the study sponsor

If the study sponsor determines to terminate or suspend the entire study, study center directors and regulatory authorities will be notified immediately in writing of this decision and reasons for it. If a study center director receives notification of termination or suspension of the study from the study sponsor, they will immediately notify in writing the investigator and IRB of this fact, including detailed reasons.

If an investigator receives notification of the termination or suspension of the study from the study center director, he or she will immediately inform subjects and ensure that appropriate medical treatments are performed.

See "12.2 Procedures for Withdrawal" for actions taken related to subjects upon study termination.

#### (3) Termination or suspension of study at a study center by investigator or IRB

If an investigator determines on his or her own judgment to terminate or suspend the study, he or she will immediately inform the study center director in writing of the details regarding this decision. The study center director will then immediately inform the study sponsor and IRB in writing.

If the IRB determines to terminate or suspend the study, it will immediately inform the study center director in writing of the details regarding this decision. The study center director will then immediately inform the investigator and study sponsor in writing.

#### (4) Termination due to dissolution of contract with study center

The study sponsor will immediately inform the regulatory authorities if it terminates the study at a study center due to serious or continued violations of GCP or the study protocol during the study period.

# 17. Case report forms

#### 17.1 Case report form (CRF) format

This study will use electronic CRFs using an electronic data capture (EDC) system. Electronic CRFs reviewed and digitally signed by investigators will be considered originals. Test results from clinical laboratory tests performed at the contract testing facility will be obtained from that facility.

# 17.2 Direct recording of information in the CRF and CRF as source documents

There is no item or category in the current study for which the electronic CRF is considered the

source document. If data from an electronic CRF is to be considered the source document, this will be agreed upon separately in writing by the study sponsor and investigator prior to initiation of the study.

# 17.3 Notes on making CRF entries

Investigators/subinvestigators or clinical coordinators will make CRF entries according to the following stipulations. CRFs will be created according to "Procedures for CRF modifications or revisions,"\* to be supplied separately by the study sponsor.

\*"Procedures for CRF modifications or revisions": eCRF operation manual and eCRF input manual

- (1) The study sponsor will perform user management duties, such as giving user names and passwords to investigators/subinvestigators and clinical research staff, which will not be shared beyond the person to which they were originally assigned. Data entry will be performed only by those with authority to do so (investigators/subinvestigators and clinical research staff).
- (2) CRFs will be created for all subjects who transitioned to the treatment period (subjects with completed treatment period enrollment).
- (3) Investigators may record any information in CRFs. Subinvestigators may record any information in CRFs excluding digital signatures. Clinical research staff may transfer information from source documents to the CRF which do not require medical judgment, such as treatment records.
- (4) When information recorded in CRFs is modified or revised, the reason for this will be recorded electronically in the CRF.
- (5) Investigators will electronically sign the CRF on the EDC system after reviewing it and confirming accuracy and completeness, and that audit trails and electronic signature information are viewable.
- (6) Investigators will retain copies of CRFs on recording media such as CDRs (stored as PDF copies of the electronic CRF after review by the investigator). Granting electronic access to CRFs (permission to view on the EDC system) may serve in lieu of submitting copies in the period from electronic signing until submission of the CDRs or other storage media.
- (7) If there is conflicting data between data in the CRF and source documents, the investigator will submit a document containing the reason for this discrepancy to the study sponsor, and retain a copy.

#### 17.4 CRF submission timepoints

Investigators/subinvestigators will make CRF entries in principle within 72 hours after each observation in the study period and after completion of evaluation, then submit these to the study

sponsor.

#### 18. Direct access to source documents

Investigators and study center directors shall grant direct access to all source documents related to the study in response to monitoring or auditing by the study sponsor, or in response to investigations by the IRB or regulatory authorities.

# 19. Study quality control and quality assurance

In order to ensure a high level of quality for the study, the study sponsor must perform study quality control and quality assurance based on Mitsubishi Tanabe Pharma Corporation's GCP procedures. Further, the contract research organization will perform study quality control based upon standard operating procedures agreed upon with the study sponsor. Meanwhile, study centers and investigators will grant their cooperation in performance of these duties.

As a part of quality control efforts, study monitors will directly observe activities as appropriate to ensure that the study is compliant with related procedures, the latest version of the study protocol, and GCP. Monitors will also confirm that information recorded in CRFs by investigators/subinvestigators can be compared with source documents and other related materials in order to verify accuracy and completeness.

The study auditor will audit the study in accordance with the GCP Standard Operating Procedure to ensure compliance with the study protocol and GCP, and otherwise confirm appropriate implementation of quality control measures.

#### 20. Ethics

# 20.1 Ethical conduct of the study

This study will be performed in accordance with the ethical principles of the Declaration of Helsinki, and in compliance with the Pharmaceutical Affairs Law, GCP, and the study protocol.

#### 20.2 Institutional Review Board

The Institutional Review Board (IRB) of each study center will review the study (including its continuation) based on the investigator's Brochure (IB), study protocol, and informed consent forms and written information for subjects from ethical, scientific, medical, and pharmaceutical perspectives.

# 20.3 Subject confidentiality

Identification of each subject through enrollment and CRFs shall be possible only with the subject identification code. All personnel involved with the current study shall endeavor to preserve subject confidentiality during direct access to source documents, publishing in academic journals, and submissions to regulatory authorities.

# 21. Record storage

#### (1) Records stored by study centers

The records storage manager appointed by each study center director shall store all study-related documents and other records to be stored at each study center until 1) or 2) below, whichever comes later. However, if the study sponsor requests that these materials be stored for a longer period, each study center will discuss storage methods and periods with the study sponsor.

If the study sponsor determines not to include materials related to results from the clinical study in the application, it will notify study center directors of this fact and the reasons for it in writing.

Further, the study sponsor will notify study center directors in writing if marketing approval is granted for the study drug, or if approval is not granted and development is canceled.

- 1) Day of marketing approval for the study drug (or 3 years from receipt of notification if notified of cancelation of development, or that study results will not be included in application)
- 2) Three years from the day of termination or completion of the study

### (2) Records stored by the study sponsor

The study sponsor shall store all study-related documents and other records to be stored by the study sponsor until 1) or 2) below, whichever comes later.

- 1) Five years from the day of marketing approval for the study drug, or day of completion of re-review (or 3 years from the date of cancellation of development)
- 2) Three years from the day of termination or completion of the study

#### 22. Monetary compensation

Monetary compensation made to study subjects and study centers will be paid in accordance with contracts and agreements between the study centers and the study sponsor.

# 23. Compensation for health damage and insurance

# 23.1 Compensation for health damage

In the event that a subject experiences damage to health related to the study, the study sponsor shall provide compensation according to determined standards (excluding instances in which causal relationship with the study has been denied). Forms of said compensation may include the subject's portion of medical coverage, treatment allowances, or financial compensation. In these events, it shall not be the burden of the subject to prove causal relationship with the study.

#### 23.2 Insurance

The study sponsor shall procure health insurance and take other measures to ensure fulfillment of liability and compensatory responsibilities to subjects related to damage to health arising from the study.

# 24. Publication policy

Information contained within this study protocol is the property of the study sponsor. Although it is provided to investigators/subinvestigators, others involved with the study, and IRBs, information contained herein shall not be disclosed to third parties without express written consent of the study sponsor, save when doing so is required for the study itself.

Information obtained through the study may be published (to academic societies, journals, etc.) by investigators/subinvestigators, or others involved with the study at study centers, only after obtaining prior consent from the study sponsor.

Finally, the study sponsor reserves the right to freely use information obtained through the study for any purpose, including reports to regulatory authorities, appropriate drug use, and sales promotions.

# 25. Genetic analysis study

# 25.1 Purpose of the study

| | Researching the relationship between genetic factors and drug efficacy as well as incidence of AEs |
|---|---|
| is | a crucial step in establishing safe, effective drugs. |

# 25.2 Eligible subjects

# 25.3 Obtaining consent

Investigators will obtain cooperation from the study sponsor in drafting informed consent forms and written information for the genetic analysis study separate from those required for the main study.

Authored or revised consent forms will be submitted to study sponsor and approved by the Institutional Review Board (IRB).

Investigators/subinvestigators will use the informed consent forms and written information for the genetic analysis study to fully explain the study to subjects and obtain their consent in writing prior to collecting blood samples for the genetic analysis study.

Investigators/subinvestigators and subjects will sign (or print name and affix personal seals to) and date these consent forms, after which subjects will receive a copy of the completed form. If clinical coordinators performed supplementary explanations, they will also sign (or print name and affix personal seal) and date the form.

Subjects may still participate in the main study even if they do not grant consent for the genetic analysis study.

# 25.4 Sample handling

### 25.4.1 Blood sampling dates

| 25.4.2 Storage an | l transport cor | aditions |
|-------------------|-----------------|----------|
|-------------------|-----------------|----------|

| Co | ollec | ted blo | od sampl | es will | be cryoj | preserve | d un | til transp | ort. The | contract 1 | testing l | laboratory | will |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| send | the | blood | samples | to the | storage | facility | for | genetic | analysis | samples. | | | |
| | | | | 11 | | | | | | | | | |

# 25.4.3 Procedures for anonymization and encoding, and preparation/storage of the identification table

The storage facility for genetic analysis samples will issue an anonymized identification number for each blood sample received, which is separate from the subject identification code. The facility will store a table linking identification codes to subjects. Methods for anonymization and creation/storage of the identity table will adhere to operating procedures of the facility or the study protocol.

# 25.4.4 Provision of the identity table

The storage facility for genetic analysis samples will provide a copy of the table linking subjects and identification codes to the study sponsor after storage of the final sample.

| | <br> |
|------|------|
| | <br> |
| D. C | |

# 25.5 Performing genetic analysis

# 25.6 Publication of results and disclosure to sample donors

#### 25.6.1 Publication of results and disclosure to sample donors

Information obtained through the genetic analysis study may be published (to academic societies, journals, etc.) by investigators/subinvestigators, or others involved with the study at study centers, only after obtaining prior consent from the study sponsor. Finally, the study sponsor reserves the right to freely use information obtained through the study for any purpose, including reports to regulatory authorities, appropriate drug use, and sales promotions.

In principle, genetic information about individual subjects will not be disclosed to either subjects themselves or study centers.

#### 25.6.2 Disposal of individual genetic information

If disposal of a sample becomes necessary due to retraction of subject consent or other reasons, the genetic information manager appointed at the time of the genetic analysis study will delete data related to the relevant subject from computers where that information is stored. Paper records will be shredded to a state where restoration is impossible. However, if retraction of consent occurs after an individual's data has already been used in a group analysis, results from that analysis may be used even after the retraction. Further, it may be impossible to fully discard results if already published in papers or other forms. Details regarding disposal of genetic information will adhere to separate procedures or study protocols to be drafted.

# 26. Administrative structure

#### 26.1 Study sponsor:

See Appendix 1.

# 26.2 Study centers and investigators

See Appendix 2.

Investigator duties: Agreeing with study protocol created by study sponsor, drafting and revising

informed consent forms and written information for subjects, selecting subjects and obtaining consent, performing study, providing medical care and information to subjects, instructing and overseeing subinvestigators and clinical coordinators, providing materials and information, cooperating with monitors and auditors, reporting deviations from the study protocol, changes from the study protocol, and AEs, making CRF entries, and storing documents or records related to the study.

### 27. References

- (1) Japanese Society of Nephrology, "Clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012." Tokyo; Tokyo Igakusha; 2012.
- (2) Iseki K. Chronic kidney disease in japan. Intern Med. 2008;47(8):681-9.
- (3) Imai E, Yasuda Y, Makino H. Japan association of chronic kidney disease initiatives (J-CKDI). Japan Med Assoc J. 2011;54(6):403-5.
- (4) Iseki K, Kohagura K. Anemia as a risk factor for chronic kidney disease. Kidney Int Suppl. 2007;(107):S4-9.
- (5) Di Iorio B, Cirillo M, Bellizzi V, Stellato D, De Santo NG; Campania Dialysis Registry Research Group. Prevalence and correlates of anaemia and uncontrolled anaemia in chronic hemodialysis patients-the Campania Dialysis Registry. Int J Artif Organs. 2007;30(4):325-33.
- (6) Stauffer ME, Fan T. Prevalence of anaemia in chronic kidney disease in the United States. PLoS One. 2014;9(1):e84943.
- (7) Nurko S. Anemia in chronic kidney disease: causes, diagnosis, treatment. Cleve Clin J Med. 2006;73(3):289-297.
- (8) Metivier F, Marchais SJ, Guerin AP, Pannier B, London GM. Pathophysiology of anaemia: focus on the heart and blood vessels. Nephrol Dial Transplant. 2000;15 Suppl 3:14-8.
- (9) National Institute for Health and Care Excellence. Chronic kidney disease: managing anaemia. NICE guideline. 2015. https://www.nice.org.uk/guidance/NG8
- (10) KDOQI; National Kidney Foundation. Clinical Practice Guidelines and Clinical Practice Recommendations for Anemia in Chronic Kidney Disease. Am J Kidney Dis. 2006;47(5 Suppl 3):S11-145.
- (11) Bigham AW, Lee FS. Human high-altitude adaptation: forward genetics meets the HIF pathway. Genes Dev. 2014;28(20):2189-204.
- (12) Committee for Statistical Survey, Japanese Society for Dialysis Therapy. The current state of dialysis treatment in Japan (as of Dec. 31, 2012). 2014;47(1):1-56.

# **Contact Information** Mitsubishi Tanabe Pharma Corporation 17-10 Nihonbashi Komai-cho, Chuo-ku, Tokyo Japan 103-8405 [Contract Monitoring Organization] Night/Holiday Contact Information Emergency contact for after-hours (between 5:30 PM and 9 AM), weekends, and holidays is given below. The call center will contact study monitors on an emergency basis.